CLINICAL TRIAL: NCT01992536
Title: Phase 2, Observer-Blind, Placebo-Controlled, Randomized, Multi-Center Extension Study to Evaluate the Safety and Immunogenicity of a Booster Dose of a MenABCWY Vaccine Administered 24 Months Following the Primary Series to Adolescents and Young Adults Who Participated in V102_03 (NCT01272180)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Vaccines (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: V102_03E1; 2012-003937-41 (EudraCT Number)
Record Dates: First submitted 2013-11-15; First posted 2013-11-25 (Estimated); Results first posted 2016-10-25 (Estimated); Last update posted 2016-10-25 (Estimated); Status verified 2016-08

CONDITIONS: Meningococcal Disease
Keywords: Meningococcal; Booster; MenABCWY; Menveo; Vaccine Adolescents; Immune Response; N. Meningitidis
MeSH Terms: conditions — Meningococcal Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (9):
- Ia: MenABCWY+OMV (Experimental): Investigational
  Interventions: Biological: MenABCWY+OMV
- Ib: Placebo (Placebo Comparator): Saline
  Interventions: Biological: Placebo
- IIa: MenABCWY+¼OMV (Experimental): Investigational
  Interventions: Biological: MenABCWY+¼OMV
- IIb: Placebo (Placebo Comparator): Saline
  Interventions: Biological: Placebo
- IIIa: MenABCWY+OMV (Experimental): Investigational
  Interventions: Biological: MenABCWY+OMV
- IIIb: MenABCWY+¼OMV (Experimental): Investigational
  Interventions: Biological: MenABCWY+¼OMV
- IVa: MenABCWY+OMV (Experimental): Investigational
  Interventions: Biological: MenABCWY+OMV
- IVb: MenABCWY+¼OMV (Experimental): Investigational
  Interventions: Biological: MenABCWY+¼OMV
- IVc: Placebo (Placebo Comparator): Saline
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: MenABCWY+OMV — Vaccine contains rMenB (50 µg per antigen) with 25 µg of OMV (a "full" dose) plus the fully lyophilized MenACWY vaccine
  Arms: IIIa: MenABCWY+OMV; IVa: MenABCWY+OMV; Ia: MenABCWY+OMV
Biological: MenABCWY+¼OMV — Vaccine contains rMenB (50 µg per antigen) with 6.25 µg OMV (1/4 dose) plus the fully lyophilized MenACWY vaccine
  Arms: IIIb: MenABCWY+¼OMV; IIa: MenABCWY+¼OMV; IVb: MenABCWY+¼OMV
Biological: Placebo — Saline solution for injection (0.5mL)
  Arms: IIb: Placebo; IVc: Placebo; Ib: Placebo

SUMMARY:
The purpose of this extension study is to evaluate the immunogenicity and safety of a booster dose of a MenABCWY vaccine, administered 24 months after completion of the primary vaccination series, in subjects who previously received the same vaccine formulation in study V102_03 (NCT01272180) (Groups I and II). Antibody persistence at 24 and 36 months after the primary vaccination and 12 months after the booster dose will also be evaluated in these subjects.

In addition, safety and immunogenicity of two investigational MenABCWY vaccine formulations (either a MenABCWY+ OMV or a MenABCWY+¼ OMV) will be assessed in subjects who previously received two doses of MenB vaccine (Group III) or one dose of Menveo vaccine (Group IV). These subjects will be followed for safety and immunogenicity for 12 months after vaccination in study V102_03E1.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females that received both vaccinations and completed the Study Termination visit in the primary study, V102_03 (NCT01272180);
2. Individuals or the individual's parents or legal guardian who have given written consent after the nature of the study has been explained according to local regulatory requirements;
3. Individuals who have given written assent as required by local regulations after the nature of the study has been explained to them according to local regulatory requirements;
4. Individuals in good health as determined by the outcome of medical history, physical examination and clinical judgment of the investigator;
5. Individuals and/or or the individual's parents or legal guardian who can comply with study procedures and are available for follow-up.

Exclusion Criteria:

1. History of any meningococcal vaccine administration other than the vaccination administered in the primary study, V102_03 (NCT01272180);
2. Current or previous, confirmed or suspected disease caused by N. meningitidis;
3. Household contact with and/or intimate exposure to an individual with any laboratory confirmed N. meningitidis infection within 60 days of enrollment;
4. History of severe allergic reactions after previous vaccinations or hypersensitivity to any vaccine component;
5. All sexually active females that have not used an "acceptable contraceptive method(s)" for at least 2 months prior to study entry. Acceptable birth control methods are defined as one or more of the following:

   1. Hormonal contraceptive (such as oral, injection, transdermal patch, implant, cervical ring)
   2. Barrier (condom with spermicide or diaphragm with spermicide) each and every time during intercourse
   3. Intrauterine device (IUD)
   4. Monogamous relationship with vasectomized partner. Partner must have been vasectomized for at least six months prior to the subject's study entry;
6. Sexually active females that refuse to use to an "acceptable contraceptive method" through to 3 weeks following the study vaccination;
7. Female subjects with a positive pregnancy test prior to the study vaccine being administered;
8. Nursing (breastfeeding) mothers;
9. Individuals with a history of illness or with an ongoing illness that, in the opinion of the investigator, may pose additional risk to the subject if he/she participates in the study;
10. Any serious, chronic, or progressive disease (e.g., neoplasm, diabetes, cardiac disease, hepatic disease, progressive neurological disease or seizure disorder; autoimmune disease, HIV infection or AIDS, blood dyscrasias, bleeding diathesis, signs of cardiac or renal failure, or severe malnutrition);
11. Subjects who required chronic administration (defined as more than 14 days) of immunosuppressants or other immune-modifying drugs within six months prior to the study vaccination. (For corticosteroids, this means prednisone, or equivalent, ≥ 20mg/day. Inhaled and topical steroids are allowed).
12. Receipt of blood, blood products and/or plasma derivatives, or a parenteral immunoglobulin preparation within the previous 90 days;
13. Individuals participating in any clinical trial with another investigational product 30 days prior to first study visit or intent to participate in another clinical study at any time during the conduct of this study;
14. Administration or planned administration, of any vaccine not foreseen by the study protocol within 30 days prior study vaccination, and up to 30 days after the vaccination (with the exception of any licensed influenza vaccine which may be administered >14 days preceding or >14 days following the study vaccination);
15. Individuals who study personnel or immediate family members of study personnel including brother, sister, child, parent, or the spouse.
16. Individuals who have experienced moderate or severe acute infection and/or fever (defined as temperature ≥ 38°C) within 3 days prior to enrolment.
17. Who have received systemic antibiotic treatment within 7 days prior to enrollment.

Ages: 10 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 194 (Actual)
Dates: Start 2013-12; Primary Completion 2014-05 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Vaccines, Study Chair — Novartis Vaccines
Locations (13):
- United States (8):
  - Site 23, Alabama Clinical Therapeutics 806 St. Vincent's Drive, Suite 615, Birmingham, Alabama
  - Site 24, Madera Family Medical Group 1111 West 4th Street, Madera, California
  - Site 25, Center for Clinical Trials LLC 16660 Paramount Blvd, Suite 301, Paramount, California
  - Site 28, Kentucky Pediatric/Adult Research 201 South 5th Street, Bardstown, Kentucky
  - Site 21, Bluegrass Clinical Research Inc. 5512 Bardstown Road, Suite 2, Louisville, Kentucky
  - Site 26, Ohio Pediatric Research Association 7200 Poe Ave, Suite 200, Dayton, Ohio
  - Site 27, Ohio Pediatric Research Association 1775 Delco Park Drive, Kettering, Ohio
  - Site 22, Focus Research Group 201 Signature Place, Lebanon, Tennessee
- Poland (5):
  - Site 15, Specjalistyczna Przychodnia Lekarska Internistyczno-Pediatryczna, Juniperus" s.c., ul.Kościuszki 41, Izabelin
  - Site 13, Hanna Czajka Indywidualna Specjalistyczna Praktyka Lekarska, Ul. Braci Kiemliczów 14, Kraków
  - Site 12, NZOZ PRAKTIMED Sp.zo.o, ul.Strzelców 15, Kraków
  - Site 14, Klinika Pediatrii Centrum Medycznego Kształcenia Podyplomowego,Szpital Bielański, Ul. Cegłowska 80, Warszawa
  - Site 11, Katedra i Klinika Pediatrii i Chorób Infekcyjnych, ul.O.Bujwida 44, Wrocław

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from 5 study sites in Poland and from 8 study sites in United States.
Pre-assignment Details: All enrolled subjects were included in the study.
Groups:
- 2OMV_OMV: Subjects who previously received two doses of MenABCWY + OMV in the parent study, received one booster dose of same vaccine in this study.
- 2OMV_Pbo: Subjects who previously received two doses of MenABCWY + OMV in the parent study, received one dose of saline solution in this study.
- 2qOMV_qOMV: Subjects who previously received two doses of MenABCWY + ¼ OMV in the parent study, received one booster dose of same vaccine in this study.
- 2qOMV_Pbo: Subjects who previously received two doses of MenABCWY + ¼ OMV in the parent study, received one dose of saline solution in this study.
- 2B_OMV: Subjects who previously received two doses of rMenB + OMV in the parent study, received one dose of MenABCWY + OMV in this study.
- 2B_qOMV: Subjects who previously received two doses of rMenB + OMV in the parent study, received one dose of MenABCWY + ¼ OMV in this study.
- 2B_Pbo: Subjects who previously received two doses of rMenB + OMV in the parent study, received one dose of Placebo in this study.
- 1M_OMV: Subjects who previously received one dose of MenACWY in the parent study, received one dose of MenABCWY + OMV in this study.
- 1M_qOMV: Subjects who previously received one dose of MenACWY in the parent study, received one dose of MenABCWY + ¼ OMV in this study.
- 1M_Pbo: Subjects who previously received one dose of MenACWY in the parent study, received one dose of saline solution in this study.
Period: Overall Study
Arm/Group | 2OMV_OMV | 2OMV_Pbo | 2qOMV_qOMV | 2qOMV_Pbo | 2B_OMV | 2B_qOMV | 2B_Pbo | 1M_OMV | 1M_qOMV | 1M_Pbo
Started | 26 | 25 | 17 | 24 | 11 | 21 | 7 | 21 | 19 | 19
Completed | 22 | 22 | 16 | 22 | 11 | 20 | 0 | 21 | 18 | 18
Not Completed | 4 | 3 | 1 | 2 | 0 | 1 | 7 | 0 | 1 | 1
Not completed — Administrative Reason | 0 | 0 | 0 | 0 | 0 | 0 | 7 | 0 | 0 | 0
Not completed — Lost to Follow-up | 4 | 2 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 1
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 2OMV_OMV | 2OMV_Pbo | 2qOMV_qOMV | 2qOMV_Pbo | 2B_OMV | 2B_qOMV | 2B_Pbo | 1M_OMV | 1M_qOMV | 1M_Pbo | Total
Number analyzed (Participants) | 26 | 25 | 17 | 24 | 11 | 21 | 7 | 21 | 19 | 19 | 190
Age, Continuous [Mean (Standard Deviation); unit: Years] | 18.8 (5.19) | 17.1 (4.31) | 18 (5.05) | 19 (5.4) | 20.9 (3.99) | 19.7 (5.36) | 17.9 (4.67) | 16.8 (4.65) | 19.2 (6.1) | 17.6 (5.19) | 18.4 (5.08)
Sex/Gender, Customized [Number; unit: Participants]
  Female | 8 | 13 | 9 | 14 | 2 | 15 | 3 | 12 | 12 | 11 | 99
  Male | 18 | 12 | 8 | 10 | 9 | 6 | 4 | 9 | 7 | 8 | 91

OUTCOME MEASURES:

1. Primary Outcome: 1. Percentages of Subjects With HT-hSBA (High-throughput Human Serum Bactericidal Assay) Seroresponse Against N. Meningitidis Serogroups A, C, W and Y.
Description: Percentages of subjects having HT-hSBA seroresponse against N. meningitidis serogroups A, C, W and Y, following administration of a booster dose of MenABCWY, in the present study, in subjects who previously received the same MenABCWY vaccine formulation in study V102_03 (NCT01272180). Seroresponse to N. meningitidis serogroups A, C, W and Y is defined as: for subjects with a pre-vaccination HT-hSBA titer < 1:4, a post-vaccination hSBA titer ≥ 1:8; for subjects with a pre-vaccination hSBA titer ≥ 1:4, an increase in hSBA titer of at least four times the pre-vaccination titer.
Time Frame: Day 30
Population: Analysis was done on FAS Day 30 (Booster) population.. All subjects in the enrolled population who were randomized, actually received the study vaccination in V102_03E1 and provided an evaluable serum sample at Day 30 (for seroresponse, Day 1 and Day 30 samples were required).
Measure: Number (95% Confidence Interval); unit: Percentages of Subjects
Arm/Group | 2OMV_OMV | 2qOMV_qOMV
Number analyzed (Participants) | 25 | 16
Percentages of Subjects
  Men A | 96 [79.6 to 99.9] | 94 [69.8 to 99.84]
  Men C (N=20,10) | 85 [62.1 to 96.8] | 100 [69.2 to 100]
  Men W (N=20,13) | 85 [62.1 to 96.8] | 85 [54.6 to 98.1]
  Men Y (N=25,14) | 96 [79.6 to 99.9] | 100 [76.8 to 100]

2. Primary Outcome: 2. Percentage of Subjects With HT-hSBA Titers ≥ 1:5 Against Strains of N. Meningitidis Serogroups B.
Description: Percentage of subjects reporting HT-hSBA titers ≥ 1:5 against strains of N. meningitidis serogroups B at baseline (Day 1) and one month (Day 30) following administration of a booster dose of MenABCWY, in the present study, in subjects who previously received the same MenABCWY vaccine formulation in study V102_03 (NCT01272180).
Time Frame: Day 1 and Day 30
Population: Analysis was done on FAS Day 30 (Booster) population. All subjects in the enrolled population who were randomized, actually received the study vaccination in V102_03E1 and provided an evaluable serum sample at Day 30 (for seroresponse, Day 1 and Day 30 samples were required).
Measure: Number (95% Confidence Interval); unit: Percentages of Subjects
Arm/Group | 2OMV_OMV | 2qOMV_qOMV
Number analyzed (Participants) | 25 | 17
Percentages of Subjects
  5/99 (Day 1, N= 25,15) | 76 [54.9 to 90.6] | 87 [59.5 to 98.3]
  5/99 (Day 30, N=25,17) | 100 [86.3 to 100.0] | 100 [80.5 to 100.0]
  H44/76 (Day 1, N=25,16) | 16 [4.5 to 36.1] | 13 [1.6 to 38.3]
  H44/76 (Day 30, N=25,17) | 96 [79.6 to 99.90] | 100 [80.5 to 100.0]
  M01-0240364 (Day 1, N=24,15) | 25 [9.8 to 46.7] | 20 [4.3 to 48.1]
  M01-0240364 (Day 30, N=25,17) | 100 [86.3 to 100.0] | 100 [80.5 to 100.0]
  M07-0241084 (Day 1,N=25,15) | 36 [18.0 to 57.5] | 27 [7.8 to 55.1]
  M07-0241084 (Day 30, N=25,17) | 100 [86.3 to 100.0] | 88 [63.6 to 98.5]
  M14459 (Day 1, N=25,15) | 24 [9.4 to 45.1] | 7 [0.17 to 31.9]
  M14459 (Day 30, N=25,17) | 92 [74.0 to 99.0] | 88 [63.6 to 98.5]
  NZ98/254 (Day 1, N=25,15) | 16 [4.5 to 36.1] | 7 [0.17 to 31.9]
  NZ98/254 (Day 30, N=25,17) | 92 [74.0 to 99.0] | 71 [44.0 to 89.7]

3. Secondary Outcome: 3. Percentage of Subjects With HT-hSBA Titer ≥ 1:8 to N. Meningitides Serogroups A, C, W, Y.
Description: Percentage of subjects with HT-hSBA titer ≥ 1:8 in serogroups A, C, W, Y against N. meningitides assessed prior to the administration of MenABCWY booster vaccination or placebo.
  Pre vaccination is 24 months after completion of the primary vaccination series, in subjects who previously received the same vaccine formulation in study V102_03 (NCT01272180).
Time Frame: Day 1 (Pre vaccination)
Population: Analysis was done on FAS Day 1 (Persistence) population. All subjects in the enrolled population who provided an evaluable serum sample at Day 1.
Measure: Number (95% Confidence Interval); unit: Percentages of Subjects
Groups:
- ABCWY+OMV: Subjects received two doses of MenABCWY + OMV administered two months apart.
- ABCWY+qOMV: Subjects received two doses of MenABCWY + qOMV administered two months apart.
- rMenB+OMV: Subjects received two doses of rMenB + OMV, administered two months apart.
- Menveo: Subjects received a dose of placebo followed by one dose of MenACWY administered two months later.
Arm/Group | ABCWY+OMV | ABCWY+qOMV | rMenB+OMV | Menveo
Number analyzed (Participants) | 51 | 40 | 38 | 59
Percentages of Subjects
  Men A (N=51,40,38,58) | 27 [15.9 to 41.7] | 28 [14.6 to 43.9] | 29 [15.4 to 45.9] | 31 [19.5 to 44.5]
  Men C (N=48,38,38,58) | 67 [51.6 to 79.6] | 68 [51.3 to 82.5] | 45 [28.6 to 61.7] | 57 [43.2 to 69.8]
  Men W (N=50,36,38,56) | 92 [80.8 to 97.8] | 75 [57.8 to 87.9] | 76 [59.8 to 88.6] | 68 [54 to 79.7]
  Men Y (N=51,38,38,59) | 65 [50.1 to 77.6] | 50 [33.4 to 66.6] | 16 [6 to 31.3] | 46 [32.7 to 59.2]

4. Secondary Outcome: 4. Percentage of Subjects With HT-hSBA Titer ≥ 1:5 to N. Meningitidis Strains of Serogroup B.
Description: Percentage of subjects with HT-hSBA titer ≥ 1:5 against N. meningitidis strains of serogroup B assessed prior to the administration of MenABCWY booster vaccination or placebo.
  Pre vaccination is 24 months after completion of the primary vaccination series, in subjects who previously received the same vaccine formulation in study V102_03 (NCT01272180).
Time Frame: Day 1 (Pre vaccination)
Population: Analysis was done on the FAS Day 1 (Persistence) population. All subjects in the enrolled population who provided an evaluable serum sample at Day 1.
Measure: Number (95% Confidence Interval); unit: Percentages of Subjects
Arm/Group | ABCWY+OMV | ABCWY+qOMV | rMenB+OMV | Menveo
Number analyzed (Participants) | 51 | 39 | 38 | 59
Percentages of Subjects
  5/99 (N=51,38,36,59) | 76 [62.5 to 87.2] | 87 [71.9 to 95.6] | 94 [81.3 to 99.3] | 19 [9.7 to 30.9]
  H44/76 (N=51,39,38,59) | 22 [11.3 to 35.3] | 18 [7.5 to 33.5] | 34 [19.6 to 51.4] | 3 [0.41 to 11.7]
  M01-0240364 (N=50,37,37,58) | 24 [13.1 to 38.2] | 16 [6.2 to 32.0] | 35 [20.2 to 52.5] | 7 [1.9 to 16.7]
  M07-0241084 (N=51,38,38,59) | 37 [24.1 to 51.9] | 29 [15.4 to 45.9] | 50 [33.4 to 66.6] | 22 [12.3 to 34.7]
  M14459 (N=51,39,38,59) | 29 [17.5 to 43.8] | 13 [4.3 to 27.4] | 26 [13.4 to 43.1] | 14 [6.0 to 25.0]
  NZ98/254 (N=51,39,38,59) | 24 [12.8 to 37.5] | 8 [1.6 to 20.9] | 16 [6.0 to 31.3] | 3 [0.41 to 11.7]

5. Secondary Outcome: 5. The HT-hSBA Geometric Mean Titers (GMTs) Against N. Meningitidis Serogroups A, C, W,Y.
Description: The HT-hSBA GMTs against N. meningitidis serogroup A, C, W, Y prior the administration of MenABCWY booster vaccination or placebo.
  Pre vaccination is 24 months after completion of the primary vaccination series, in subjects who previously received the same vaccine formulation in study V102_03 (NCT01272180).
Time Frame: Day 1 (Pre-vaccination)
Population: as for outcome 3
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | ABCWY+OMV | ABCWY+qOMV | rMenB+OMV | Menveo
Number analyzed (Participants) | 51 | 40 | 38 | 59
Titers
  Men A (N=51,40,38,58) | 3.34 [2.19 to 5.08] | 3.3 [1.95 to 5.60] | 2.96 [1.70 to 5.17] | 4.14 [2.75 to 6.23]
  Men C (N=48,38,38,58) | 18 [11 to 30] | 13 [8.00 to 20] | 6.05 [4.28 to 8.55] | 10 [6.36 to 17]
  Men W (N=50,36,38,56) | 35 [24 to 52] | 23 [12 to 45] | 20 [11 to 34] | 17 [9.65 to 29]
  Men Y (N=51,38,38,59) | 13 [7.01 to 23] | 8.85 [4.24 to 18] | 1.8 [1.25 to 2.60] | 6.49 [3.72 to 11]

6. Secondary Outcome: 6. The HT-hSBA GMTs Against N. Meningitidis Strains of Serogroup B.
Description: The HT-hSBA GMTs against N. meningitidis strains of serogroup B prior the administration of MenABCWY booster vaccination or placebo.
  Pre vaccination is 24 months after completion of the primary vaccination series, in subjects who previously received the same vaccine formulation in study V102_03 (NCT01272180).
Time Frame: Day 1 (Pre-vaccination)
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | ABCWY+OMV | ABCWY+qOMV | rMenB+OMV | Menveo
Number analyzed (Participants) | 50 | 38 | 36 | 17
Titers
  5/99 (N=51,38,36,59) | 16 [11 to 24] | 33 [19 to 54] | 39 [25 to 62] | 2.46 [1.73 to 3.51]
  H44/76 (N=51,39,38,59) | 2.54 [1.69 to 3.82] | 1.78 [1.26 to 2.53] | 3.22 [2.18 to 4.76] | 1.32 [1.06 to 1.65]
  M01-0240364 (N=50,37,37,58) | 2.67 [1.70 to 4.20] | 2.1 [1.21 to 3.65] | 4.72 [2.44 to 9.13] | 1.37 [1.06 to 1.78]
  M07-0241084 (N=51,38,38,59) | 3.76 [2.55 to 5.56] | 2.42 [1.70 to 3.45] | 4.56 [2.97 to 7.01] | 2.35 [1.68 to 3.28]
  M14459 (N=51,39,38,59) | 2.67 [1.92 to 3.70] | 1.94 [1.48 to 2.56] | 2.82 [2.00 to 3.96] | 1.87 [1.43 to 2.43]
  NZ98/254 (N=51,39,38,59) | 2.03 [1.43 to 2.89] | 1.46 [1.15 to 1.85] | 1.75 [1.24 to 2.47] | 1.16 [1.00 to 1.34]

7. Secondary Outcome: 7. The HT-hSBA GMTs Against N. Meningitidis Serogroups A, C, W, Y.
Description: The HT-hSBA GMTs against N. meningitidis serogroup A, C, W, Y at Day 1 and Day 30 (one month) after the administration of MenABCWY booster vaccination or placebo.
Time Frame: Day 1 and Day 30
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Groups:
- 2B_qOMV: Subjects who previously received two doses of rMenB + OMV in the parent study, received one dose of MenABCWY + ¼OMV in this study
- 1M_qOMV: Subjects who previously received one dose of MenACWY in the parent study, received one dose of MenABCWY + ¼OMV in this study.
Arm/Group | 2OMV_OMV | 2OMV_Pbo | 2qOMV_qOMV | 2qOMV_Pbo | 2B_OMV | 2B_qOMV | 1M_OMV | 1M_qOMV | 1M_Pbo
Number analyzed (Participants) | 25 | 25 | 16 | 23 | 11 | 21 | 21 | 18 | 18
Titers
  Men A (Day 1, N=25,25,16,22,11,21,19,16,18) | 3.41 [1.87 to 6.22] | 2.92 [1.59 to 5.36] | 2.86 [1.23 to 6.63] | 2.73 [1.41 to 5.27] | 2.26 [0.96 to 5.31] | 3.94 [1.58 to 9.85] | 6.62 [2.85 to 15] | 2.09 [1.28 to 3.41] | 5.02 [2.06 to 12]
  Men A (Day 30, N=25,25,16,22,11,21,19,17,18) | 259 [174 to 383] | 4.28 [2.03 to 9.03] | 333 [199 to 559] | 3.07 [1.51 to 6.25] | 438 [287 to 670] | 416 [198 to 871] | 138 [84 to 229] | 46 [24 to 87] | 4.91 [2.00 to 12]
  Men C (Day 1, N=20,23,10,22,7,16,21,18,17) | 23 [9.45 to 57] | 16 [7.06 to 36] | 17 [5.98 to 51] | 11 [6.24 to 19] | 5.45 [2.41 to 12] | 9.02 [5.24 to 16] | 7.75 [4.19 to 14] | 7.53 [2.38 to 24] | 17 [6.60 to 44]
  Men C (Day 30, N=21,24,11,23,7,16,21,18,18) | 660 [401 to 1084] | 17 [7.60 to 38] | 612 [245 to 1524] | 11 [5.51 to 22] | 292 [75 to 1142] | 135 [69 to 261] | 338 [205 to 558] | 304 [124 to 742] | 20 [7.20 to 56]
  Men W (Day 1, N=20,24,13,21,11,19,18,17,15) | 34 [20 to 59] | 33 [17 to 65] | 30 [8.90 to 101] | 18 [7.30 to 46] | 25 [7.98 to 79] | 29 [13 to 64] | 28 [12 to 66] | 9.37 [2.85 to 31] | 9.42 [3.03 to 29]
  Men W (Day 30, N=20,24,16,22,11,19,19,17,16) | 792 [516 to 1216] | 34 [16 to 71] | 880 [671 to 1154] | 26 [11 to 59] | 392 [252 to 610] | 363 [278 to 473] | 629 [384 to 1032] | 364 [180 to 736] | 16 [4.87 to 53]
  Men Y (Day 1, N=25,25,14,22,11,21,21,18,18) | 10 [4.89 to 21] | 15 [5.50 to 43] | 15 [4.33 to 53] | 5.66 [2.25 to 14] | 2.4 [1.05 to 5.47] | 1.84 [1.07 to 3.14] | 6.43 [2.86 to 14] | 5.79 [1.77 to 19] | 5.32 [1.81 to 16]
  Men Y (Day 30, N=25,25,16,23,11,21,21,18,18) | 464 [294 to 734] | 16 [5.65 to 48] | 697 [435 to 1116] | 5.17 [2.16 to 12] | 48 [14 to 157] | 39 [13 to 120] | 658 [431 to 1003] | 419 [217 to 809] | 6.36 [1.91 to 21]

8. Secondary Outcome: 8. The HT-hSBA GMTs Against N. Meningitidis Strains of Serogroups B.
Description: The HT-hSBA GMTs against N. meningitidis strains of serogroups B at Day 1 and Day 30 (one month) after the administration of MenABCWY booster vaccination or placebo.
Time Frame: Day 1 and Day 30
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | 2OMV_OMV | 2OMV_Pbo | 2qOMV_qOMV | 2qOMV_Pbo | 2B_OMV | 2B_qOMV | 1M_OMV | 1M_qOMV | 1M_Pbo
Number analyzed (Participants) | 25 | 25 | 17 | 23 | 11 | 21 | 21 | 19 | 18
Titers
  5/99 (Day 1, N=25,25,15,22,9,21,21,19,18) | 17 [9.56 to 29] | 16 [8.32 to 30] | 35 [14 to 92] | 30 [15 to 60] | 27 [8.61 to 86] | 43 [24 to 77] | 2.97 [1.58 to 5.59] | 1.74 [1.01 to 3.03] | 2.81 [1.30 to 6.06]
  5/99 (Day 30, N=25,25,17,23,11,21,21,19,18) | 1131 [716 to 1787] | 20 [10 to 42] | 1598 [900 to 2840] | 34 [20 to 59] | 2205 [1560 to 3117] | 2576 [1716 to 3867] | 28 [11 to 67] | 30 [11 to 78] | 3.41 [1.20 to 9.73]
  H44/76 (Day 1, N= 25,25,16,22,11,21,19,19,18) | 2.92 [1.50 to 5.67] | 2.03 [1.23 to 3.34] | 1.46 [0.96 to 2.21] | 1.92 [1.11 to 3.32] | 3.45 [1.81 to 6.57] | 3.24 [1.76 to 5.94] | 1.09 [0.96 to 1.22] | 1.47 [0.92 to 2.36] | 1.18 [0.97 to 1.44]
  H44/76 (Day 30, 25,25,17,23,11,21,19,19,18) | 97 [60 to 157] | 2.36 [1.39 to 4.01] | 56 [32 to 97] | 2.54 [1.42 to 4.53] | 132 [64 to 271] | 79 [42 to 149] | 5.27 [2.54 to 11] | 3.85 [1.85 to 8.02] | 1.63 [0.75 to 3.52]
  M01-0240364 (Day 1, N=24,25,15,20,10,21,20,18,18) | 2.28 [1.3 to 3.98] | 3.11 [1.44 to 6.68] | 2.67 [0.87 to 8.24] | 1.36 [0.83 to 2.23] | 2.46 [0.72 to 8.4] | 6.81 [2.47 to 19] | 1.34 [0.84 to 2.13] | 1.23 [0.88 to 1.71] | 1.63 [0.86 to 3.11]
  M01-0240364 (Day 30, N=25,25,17,22,11,21,20,19,18) | 685 [397 to 1182] | 3.21 [1.4 to 7.37] | 856 [454 to 1614] | 1.94 [1.02 to 3.69] | 1336 [810 to 2202] | 1275 [794 to 2048] | 3.5 [1.32 to 9.3] | 3.42 [1.19 to 9.8] | 1.76 [0.75 to 4.09]
  M07-0241084 (Day 1, N= 25,25,15,22,11,21,21,19,18) | 3.53 [2.09 to 5.95] | 3.54 [1.98 to 6.31] | 2.16 [1.15 to 4.08] | 2.52 [1.58 to 4.03] | 4.10 [1.89 to 8.90] | 6.08 [3.18 to 12] | 2.08 [1.26 to 3.42] | 2.06 [1.13 to 3.77] | 3.01 [1.38 to 6.56]
  M07-0241084 (Day 30, N=25,25,17,23,11,21,21,19,18) | 50 [31 to 79] | 3.66 [2.02 to 6.64] | 29 [14 to 58] | 2.48 [1.55 to 3.96] | 68 [33 to 142] | 69 [36 to 129] | 3.26 [1.75 to 6.06] | 2.15 [1.13 to 4.07] | 3.86 [1.40 to 11]
  M14459 (Day 1, N=25,25,15,23,11,21,20,19,18) | 2.57 [1.57 to 4.22] | 2.58 [1.62 to 4.12] | 1.6 [0.97 to 2.65] | 2.27 [1.61 to 3.2] | 3.11 [1.74 to 5.56] | 3.18 [1.87 to 5.41] | 1.91 [1.14 to 3.2] | 1.45 [1.03 to 2.05] | 2.37 [1.31 to 4.29]
  M14459 (Day 30, N=25,25,17,23,11,21,20,19,18) | 31 [18 to 54] | 2.18 [1.39 to 3.42] | 20 [11 to 37] | 2.33 [1.62 to 3.35] | 56 [27 to 117] | 35 [21 to 58] | 3.44 [2.05 to 5.75] | 2.57 [1.51 to 4.37] | 2.93 [1.14 to 7.53]
  NZ98/254 (Day 1, N= 25,25,15,23,11,21,21,19,18) | 1.65 [1.09 to 2.48] | 2.11 [1.28 to 3.49] | 1.32 [0.94 to 1.84] | 1.58 [1.11 to 2.27] | 1.72 [0.99 to 2.98] | 2.07 [1.17 to 3.66] | 1.18 [0.84 to 1.66] | 1.18 [0.90 to 1.54] | 1.12 [0.94 to 1.34]
  NZ98/254 (Day 30, N= 25,25,17,23,11,21,21,19,18) | 29 [18 to 47] | 2.03 [1.21 to 3.40] | 12 [5.04 to 31] | 1.87 [1.11 to 3.16] | 17 [6.22 to 45] | 28 [17 to 44] | 2.48 [1.31 to 4.69] | 1.58 [0.96 to 2.59] | 1.71 [0.84 to 3.50]

9. Secondary Outcome: 9. Percentage of Subjects With Four-fold Rise in HT-hSBA Titers Against N. Meningitidis Serogroup B Strains.
Description: Percentage of subjects with four-fold rise in HT-hSBA titers against N. meningitidis serogroup B strains, from Day 1 (baseline) to Day 30 (one month) after the administration of MenABCWY booster vaccination or placebo.
  Four-fold rise is defined as follows: for subjects with a pre-vaccination titer < 1:2, a post-titer of ≥ 1:8; for subjects with a pre-vaccination titer ≥ 1:2 at least a four-fold increase.
Time Frame: Day 1 and Day 30
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentages of Subjects
Arm/Group | 2OMV_OMV | 2OMV_Pbo | 2qOMV_qOMV | 2qOMV_Pbo | 2B_OMV | 2B_qOMV | 1M_OMV | 1M_qOMV | 1M_Pbo
Number analyzed (Participants) | 25 | 25 | 16 | 22 | 11 | 21 | 21 | 19 | 18
Percentages of Subjects
  5/99 (Day 1, N= 24,24,16,22,11,20,6,5,5) | 96 [78.9 to 99.89] | 100 [85.8 to 100.0] | 94 [69.8 to 99.84] | 100 [84.6 to 100.0] | 91 [58.7 to 99.77] | 95 [75.1 to 99.87] | 0 [0 to 45.9] | 0 [0.0 to 52.2] | 0 [0.0 to 52.2]
  5/99 (Day 30, N=25,25,15,22,9,21,21,19,18) | 100 [86.3 to 100.0] | 4 [0.10 to 20.4] | 93 [68.1 to 99.83] | 0 [0.0 to 15.4] | 100 [66.4 to 100.0] | 95 [76.2 to 99.88] | 57 [34.0 to 78.2] | 79 [54.4 to 93.9] | 6 [0.14 to 27.3]
  H44/76 (Day 1, N=24,25,16,23,11,20,6,5,5) | 100 [85.8 to 100.0] | 96 [79.6 to 99.90] | 100 [79.4 to 100.0] | 96 [78.1 to 99.89] | 91 [58.7 to 99.77] | 90 [68.3 to 98.8] | 0 [0.0 to 45.9] | 0 [0.0 to 52.2] | 0 [0.0 to 52.2]
  H44/76 (Day 30, N=25,25,16,22,11,21,19,19,18) | 84 [63.9 to 95.5] | 4 [0.10 to 20.4] | 94 [69.8 to 99.84] | 0 [0.0 to 15.4] | 100 [71.5 to 100.0] | 76 [52.8 to 91.8] | 37 [16.3 to 61.6] | 26 [9.1 to 51.2] | 6 [0.14 to 27.3]
  M01-0240364 (Day 1, N=23,23,16,20,11,20,6,5,4) | 78 [56.3 to 92.5] | 74 [51.6 to 89.8] | 63 [35.4 to 84.8] | 75 [50.9 to 91.3] | 82 [48.2 to 97.7] | 85 [62.1 to 96.8] | 0 [0.0 to 45.9] | 0 [0.0 to 52.2] | 0 [0.0 to 60.2]
  M01-0240364 (Day30,N=24,25,15,20,10,21,20,18,18) | 100 [85.8 to 100.0] | 4 [0.10 to 20.4] | 93 [68.1 to 99.83] | 5 [0.13 to 24.9] | 100 [69.2 to 100.0] | 90 [69.6 to 98.8] | 20 [5.7 to 43.7] | 22 [6.4 to 47.6] | 6 [0.14 to 27.3]
  M07-0241084 (Day 1, N=24,23,16,21,11,20,6,5,4) | 25 [9.8 to 46.7] | 17 [5.0 to 38.8] | 31 [11.0 to 58.7] | 19 [5.4 to 41.9] | 45 [16.7 to 76.6] | 55 [31.5 to 76.9] | 0 [0.0 to 45.9] | 0 [0.0 to 52.2] | 0 [0.0 to 60.2]
  M07-0241084 (Day 30,N=25,25,15,22,11,21,21,19,18) | 76 [54.9 to 90.6] | 0 [0.0 to 13.7] | 87 [59.5 to 98.3] | 0 [0.0 to 15.4] | 82 [48.2 to 97.7] | 62 [38.4 to 81.9] | 14 [3.0 to 36.3] | 0 [0.0 to 17.6] | 6 [0.14 to 27.3]
  M14459 (Day 1, N=24,25,16,22,11,20,6,5,5) | 54 [32.8 to 74.4] | 48 [27.8 to 68.7] | 63 [35.4 to 84.8] | 59 [36.4 to 79.3] | 91 [58.7 to 99.77] | 60 [36.1 to 80.9] | 0 [0.0 to 45.9] | 0 [0.0 to 52.2] | 0 [0.0 to 52.2]
  M14459 (Day 30, N=25,25,15,23,11,21,5,20,19,18) | 72 [50.6 to 87.9] | 0 [0.0 to 13.7] | 87 [59.5 to 98.3] | 0 [0.0 to 14.8] | 100 [71.5 to 100.0] | 76 [52.8 to 91.8] | 15 [3.2 to 37.9] | 5 [0.13 to 26.0] | 6 [0.14 to 27.3]
  NZ98/254 (Day 1, N=24,24,16,22,11,20,6,5,5) | 50 [29.1 to 70.9] | 46 [25.6 to 67.2] | 50 [24.7 to 75.3] | 59 [36.4 to 79.3] | 55 [23.4 to 83.3] | 70 [45.7 to 88.1] | 0 [0.0 to 45.9] | 0 [0.0 to 52.2] | 0 [0.0 to 52.2]
  NZ98/254 (Day 30, N=25,25,15,23,11,21,21,19,18) | 76 [54.9 to 90.6] | 0 [0.0 to 13.7] | 67 [38.4 to 88.2] | 4 [0.11 to 21.9] | 82 [48.2 to 97.7] | 67 [43.0 to 85.4] | 19 [5.4 to 41.9] | 5 [0.13 to 26.0] | 6 [0.14 to 27.3]

10. Secondary Outcome: 10. Percentage of Subjects With HT-hSBA Titer ≥ 1:8 Against N. Meningitidis Serogroups A,C,W,Y.
Description: Percentage of subjects with HT-hSBA titer ≥ 1:8 to N. meningitidis serogroups A,C,W,Y at Day 1 and Day 30 (one month) after the administration of a booster dose of MenABCWY vaccine or placebo in this study, versus baseline.
Time Frame: Day 1 and Day 30
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentages of Subjects
Arm/Group | 2OMV_OMV | 2OMV_Pbo | 2qOMV_qOMV | 2qOMV_Pbo | 2B_OMV | 2B_qOMV | 1M_OMV | 1M_qOMV | 1M_Pbo
Number analyzed (Participants) | 25 | 25 | 16 | 23 | 11 | 21 | 21 | 18 | 18
Percentages of Subjects
  Men A (Day 1, N=25,25,16,22,11,21,19,16,18) | 32 [14.9 to 53.5] | 20 [6.8 to 40.7] | 19 [4.0 to 45.6] | 27 [10.7 to 50.2] | 27 [6.0 to 61.0] | 33 [14.6 to 57.0] | 47 [24.4 to 71.1] | 6 [0.16 to 30.2] | 39 [17.3 to 64.3]
  Men A (Day 30, N=25,25,16,22,11,21,19,17,18) | 100 [86.3 to 100] | 36 [18 to 57.5] | 100 [79.4 to 100] | 27 [10.7 to 50.2] | 100 [71.5 to 100] | 95 [76.2 to 99.88] | 100 [82.4 to 100] | 94 [71.3 to 99.85] | 39 [17.3 to 64.3]
  Men C (Day 1, N=20,23,10,22,7,16,21,18,17) | 70 [45.7 to 88.1] | 65 [42.7 to 83.6] | 70 [34.8 to 93.3] | 68 [45.1 to 86.1] | 43 [9.9 to 81.6] | 63 [35.4 to 84.8] | 57 [34 to 78.2] | 44 [21.5 to 69.2] | 65 [38.3 to 85.8]
  Men C (Day 30, N=21,24,11,23,7,16,21,18,18) | 100 [83.9 to 100] | 63 [40.6 to 81.2] | 100 [71.5 to 100] | 61 [38.5 to 80.3] | 100 [59 to 100] | 100 [79.4 to 100] | 100 [83.9 to 100] | 89 [65.3 to 98.6] | 61 [35.7 to 82.7]
  Men W (Day 1, N=20,24,13,21,11,19,18,17,15) | 95 [75.1 to 99.87] | 88 [67.6 to 97.3] | 77 [46.2 to 95] | 71 [47.8 to 88.7] | 82 [48.2 to 97.7] | 79 [54.4 to 93.9] | 83 [58.6 to 96.4] | 53 [27.8 to 77] | 53 [26.6 to 78.7]
  Men W (Day 30, N=20,24,16,22,11,19,19,17,16) | 100 [83.2 to 100] | 79 [57.8 to 92.9] | 100 [79.4 to 100] | 77 [54.6 to 92.9] | 100 [71.5 to 100] | 100 [82.4 to 100] | 100 [82.4 to 100] | 100 [80.5 to 100] | 63 [35.4 to 84.8]
  Men Y (Day 1, N=25,25,14,22,11,21,21,18,18) | 64 [42.5 to 82] | 64 [42.5 to 82] | 64 [35.1 to 87.2] | 41 [20.7 to 63.6] | 36 [10.9 to 69.2] | 10 [1.2 to 30.4] | 52 [29.8 to 74.3] | 39 [17.3 to 64.3] | 39 [17.3 to 64.3]
  Men Y (Day 30, N=25,25,16,23,11,21,21,18,18) | 100 [86.3 to 100] | 60 [38.7 to 78.9] | 100 [79.4 to 100] | 39 [19.7 to 61.5] | 82 [48.2 to 97.7] | 76 [52.8 to 91.8] | 100 [83.9 to 100] | 100 [81.5 to 100] | 39 [17.3 to 64.3]

11. Secondary Outcome: 11. Percentage of Subjects With HT-hSBA Titer ≥ 1:5 Against N. Meningitidis Serogroup B Strains.
Description: Percentage of subjects with HT-hSBA titer ≥ 1:5 to N. meningitidis serogroup B strains at Day 1 and Day 30 (one month) after the administration of a booster dose of MenABCWY vaccine or placebo in this study, versus baseline.
Time Frame: Day 1 and Day 30
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentages of Subjects
Arm/Group | 2OMV_OMV | 2OMV_Pbo | 2qOMV_qOMV | 2qOMV_Pbo | 2B_OMV | 2B_qOMV | 1M_OMV | 1M_qOMV | 1M_Pbo
Number analyzed (Participants) | 25 | 25 | 17 | 23 | 11 | 21 | 21 | 19 | 18
Percentages of Subjects
  5/99 (Day 1, N=25,25,15,22,9,21,21,19,18) | 76 [54.9 to 90.6] | 76 [54.9 to 90.6] | 87 [59.5 to 98.3] | 86 [65.1 to 97.1] | 89 [51.8 to 99.72] | 95 [76.2 to 99.88] | 19 [5.4 to 41.9] | 16 [3.4 to 39.6] | 22 [6.4 to 47.6]
  5/99 (Day 30, N=25,25,17,23,11,21,21,19,18) | 100 [86.3 to 100] | 84 [63.9 to 95.5] | 100 [80.5 to 100] | 91 [72 to 98.6] | 100 [71.5 to 100] | 100 [83.9 to 100] | 76 [52.8 to 91.8] | 84 [60.4 to 96.6] | 22 [6.4 to 47.6]
  H44/76 (Day 1, N=25,25,16,22,11,21,19,19,18) | 16 [4.5 to 36.1] | 24 [9.4 to 45.1] | 13 [1.6 to 38.3] | 18 [5.2 to 40.3] | 45 [16.7 to 76.6] | 29 [11.3 to 52.2] | 0 [0 to 17.6] | 5 [0.13 to 26.0] | 0 [0 to 18.5]
  H44/76 (Day 30, N=25,25,17,23,11,21,19,19,18) | 96 [79.6 to 99.90] | 24 [9.4 to 45.1] | 100 [80.5 to 100] | 26 [10.2 to 48.4] | 100 [71.5 to 100] | 100 [83.9 to 100] | 58 [33.5 to 79.7] | 32 [12.6 to 56.6] | 6 [0.14 to 27.3]
  M01-0240364 (Day 1, N=24,25,15,20,10,21,20,18,18) | 25 [9.8 to 46.7] | 24 [9.4 to 45.1] | 20 [4.3 to 48.1] | 5 [0.13 to 24.9] | 20 [2.5 to 55.6] | 43 [21.8 to 66] | 5 [0.13 to 24.9] | 6 [0.14 to 27.3] | 11 [1.4 to 34.7]
  M01-0240364 (Day 30, N=25,25,17,22,11,21,20,19,18) | 100 [86.3 to 100] | 24 [9.4 to 45.1] | 100 [80.5 to 100] | 18 [5.2 to 40.3] | 100 [71.5 to 100] | 100 [83.9 to 100] | 25 [8.7 to 49.1] | 26 [9.1 to 51.2] | 11 [1.4 to 34.7]
  M07-0241084 (Day 1,N=25,25,15,22,11,21,21,19,18) | 36 [18.0 to 57.5] | 36 [18.0 to 57.5] | 27 [7.8 to 55.1] | 27 [10.7 to 50.2] | 64 [30.8 to 89.1] | 52 [29.8 to 74.3] | 19 [5.4 to 41.9] | 16 [3.4 to 39.6] | 33 [13.3 to 59.0]
  M07-0241084 (Day 30,N=25,25,17,23,11,21,21,19,18) | 100 [86.3 to 100] | 40 [21.1 to 61.3] | 88 [63.6 to 98.5] | 30 [13.2 to 52.9] | 91 [58.7 to 99.77] | 95 [76.2 to 99.88] | 33 [14.6 to 57.0] | 21 [6.1 to 45.6] | 33 [13.3 to 59.0]
  M14459 (Day 1, N=25,25,15,23,11,21,20,19,18) | 24 [9.4 to 45.1] | 32 [14.9 to 53.5] | 7 [0.17 to 31.9] | 17 [5.0 to 38.8] | 36 [10.9 to 69.2] | 29 [11.3 to 52.2] | 10 [1.2 to 31.7] | 11 [1.3 to 33.1] | 22 [6.4 to 47.6]
  M14459 (Day 30, N=25,25,17,23,11,21,20,19,18) | 92 [74 to 99] | 28 [12.1 to 49.4] | 88 [63.6 to 98.5] | 30 [13.2 to 52.9] | 100 [71.5 to 100] | 95 [76.2 to 99.88] | 35 [15.4 to 59.2] | 32 [12.6 to 56.6] | 22 [6.4 to 47.6]
  NZ98/254 (Day 1, N=25,25,15,23,11,21,21,19,18) | 16 [4.5 to 36.1] | 28 [12.1 to 49.4] | 7 [0.17 to 31.9] | 9 [1.1 to 28] | 9 [0.23 to 41.3] | 24 [8.2 to 47.2] | 5 [0.12 to 23.8] | 5 [0.13 to 26] | 0 [0 to 18.5]
  NZ98/254 (Day 30, N=25,25,17,23,11,21,21,19,18) | 92 [74 to 99] | 20 [6.8 to 40.7] | 71 [44 to 89.7] | 13 [2.8 to 33.6] | 82 [48.2 to 97.7] | 95 [76.2 to 99.88] | 19 [5.4 to 41.9] | 16 [3.4 to 39.6] | 6 [0.14 to 27.3]

12. Secondary Outcome: 12. Percentage of Subjects With Seroresponse to N. Meningitidis Serogroups A, C, W and Y, at Day 30 After Booster Vaccination in This Study.
Description: Percentage of subjects with seroresponse to N. meningitidis serogroup A, C, W and Y, at Day 30 after the administration of a booster dose of MenABCWY vaccine or placebo in this study, versus baseline.
Time Frame: Day 30
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentages of Subjects
Arm/Group | 2OMV_OMV | 2OMV_Pbo | 2qOMV_qOMV | 2qOMV_Pbo | 2B_OMV | 2B_qOMV | 1M_OMV | 1M_qOMV | 1M_Pbo
Number analyzed (Participants) | 25 | 25 | 16 | 22 | 11 | 21 | 21 | 18 | 18
Percentages of Subjects
  Men A Overall | 96 [79.6 to 99.90] | 12 [2.5 to 31.2] | 94 [69.8 to 99.84] | 0 [0 to 15.4] | 100 [71.5 to 100.0] | 86 [63.7 to 97] | 84 [60.4 to 96.6] | 94 [69.8 to 99.84] | 0 [0 to 18.5]
  Men C Overall | 85 [62.1 to 96.8] | 4 [0.11 to 21.9] | 100 [69.2 to 100.0] | 0 [0 to 15.4] | 100 [59.0 to 100.0] | 81 [54.4 to 96.0] | 95 [76.2 to 99.88] | 78 [52.4 to 93.6] | 6 [0.15 to 28.7]
  Men W Overall | 85 [62.1 to 96.8] | 4 [0.11 to 21.1] | 85 [54.6 to 98.1] | 5 [0.12 to 23.8] | 82 [48.2 to 97.7] | 68 [43.4 to 87.4] | 83 [58.6 to 96.4] | 76 [50.1 to 93.2] | 20 [4.3 to 48.1]
  Men Y Overall | 96 [79.6 to 99.9] | 4 [0.1 to 20.4] | 100 [76.8 to 100.0] | 0 [0 to 15.4] | 73 [39 to 94] | 62 [38.4 to 81.9] | 95 [76.2 to 99.88] | 89 [65.3 to 98.6] | 6 [0.14 to 27.3]

13. Secondary Outcome: 13. Percentage of Subjects With HT-hSBA Titer ≥ 1:8 to N. Meningitidis Serogroups A, C, W,Y.
Description: Percentage of subjects with HT-hSBA titer ≥ 1:8 against N. meningitidis serogroups A, C, W, Y, at 24 and 36 months after the primary vaccination.
Time Frame: Day 1 and Day 365
Population: Analysis was done on the FAS Day 365 (Persistence of Booster) population. All subjects in the enrolled population who were randomized, actually received the study vaccination in V102_03E1 and provided an evaluable serum sample at Day 365.
Measure: Number (95% Confidence Interval); unit: Percentages of Subjects
Arm/Group | 2OMV_OMV | 2OMV_Pbo | 2qOMV_qOMV | 2qOMV_Pbo | 2B_OMV | 2B_qOMV | 1M_OMV | 1M_qOMV | 1M_Pbo
Number analyzed (Participants) | 21 | 22 | 16 | 20 | 11 | 20 | 20 | 18 | 17
Percentages of Subjects
  Men A (Day 1, N= 21,22,15,20,10,20,20,17,17) | 38 [18.1 to 61.6] | 18 [5.2 to 40.3] | 20 [4.3 to 48.1] | 30 [11.9 to 54.3] | 30 [6.7 to 65.2] | 35 [15.4 to 59.2] | 45 [23.1 to 68.5] | 12 [1.5 to 36.4] | 41 [18.4 to 67.1]
  Men A (Day 365, N= 21,22,16,20,10,20,20,18,17) | 67 [43.0 to 85.4] | 23 [7.8 to 45.4] | 88 [61.7 to 98.4] | 25 [8.7 to 49.1] | 90 [55.5 to 99.75] | 85 [62.1 to 96.8] | 85 [62.1 to 96.8] | 50 [26.0 to 74.0] | 35 [14.2 to 61.7]
  Men C (Day 1, N= 20,19,14,20,11,19,19,18,16) | 65 [40.8 to 84.6] | 68 [43.4 to 87.4] | 71 [41.9 to 91.6] | 65 [40.8 to 84.6] | 36 [10.9 to 69.2] | 58 [33.5 to 79.7] | 58 [33.5 to 79.7] | 50 [26 to 74] | 75 [47.6 to 92.7]
  Men C (Day 365, N= 21,21,16,20,11,19,19,18,17) | 100 [83.9 to 100] | 62 [38.4 to 81.9] | 100 [79.4 to 100] | 50 [27.2 to 72.8] | 82 [48.2 to 97.7] | 95 [74 to 99.87] | 100 [82.4 to 100] | 89 [65.3 to 98.6] | 65 [38.3 to 85.8]
  Men W (Day 1, N= 20,22,12,20,11,20,17,18,16) | 95 [75.1 to 99.87] | 95 [77.2 to 99.88] | 75 [42.8 to 94.5] | 70 [45.7 to 88.1] | 82 [48.2 to 97.7] | 75 [50.9 to 91.3] | 82 [56.6 to 96.2] | 61 [35.7 to 82.7] | 56 [29.9 to 80.2]
  Men W (Day 365, N= 21,22,16,20,11,20,19,18,17) | 100 [83.9 to 100] | 82 [59.7 to 94.8] | 100 [79.4 to 100] | 65 [40.8 to 84.6] | 91 [58.7 to 99.77] | 100 [83.2 to 100] | 100 [82.4 to 100] | 100 [81.5 to 100] | 65 [38.3 to 85.8]
  Men Y (Day 1, N= 21,21,14,20,11,18,20,18,17) | 62 [38.4 to 81.9] | 62 [38.4 to 81.9] | 71 [41.9 to 91.6] | 40 [19.1 to 63.9] | 36 [10.9 to 69.2] | 11 [1.4 to 34.7] | 55 [31.5 to 76.9] | 44 [21.5 to 69.2] | 41 [18.4 to 67.1]
  Men Y (Day 365, N= 21,21,16,20,11,18,20,18,17) | 95 [76.2 to 99.88] | 52 [29.8 to 74.3] | 100 [79.4 to 100] | 40 [19.1 to 63.9] | 45 [16.7 to 76.6] | 72 [46.5 to 90.3] | 100 [83.2 to 100] | 89 [65.3 to 98.6] | 47 [23 to 72.2]

14. Secondary Outcome: 14. Percentage of Subjects With HT-hSBA Titer ≥ 1:5 to N. Meningitidis Strains of Serogroup B
Description: Percentage of subjects with HT-hSBA titer ≥ 1:5 against N. meningitidis strains of serogroup B, at 24 and 36 months after the primary vaccination.
Time Frame: Day 1, Day 30 and Day 365
Population: Analysis was done on FAS Day 365 (Persistence of Booster) population. All subjects in the enrolled population who were randomized, actually received the study vaccination in V102_03E1 and provided an evaluable serum sample at Day 365.
Measure: Number (95% Confidence Interval); unit: Percentages of Subjects
Arm/Group | 2OMV_OMV | 2OMV_Pbo | 2qOMV_qOMV | 2qOMV_Pbo | 2B_OMV | 2B_qOMV | 1M_OMV | 1M_qOMV | 1M_Pbo
Number analyzed (Participants) | 21 | 22 | 16 | 20 | 11 | 20 | 21 | 18 | 17
Percentages of Subjects
  5/99 (Day 1, N=21,22,14,20,9,19,21,18,17) | 76 [52.8 to 91.8] | 82 [59.7 to 94.8] | 86 [57.2 to 98.2] | 85 [62.1 to 96.8] | 89 [51.8 to 99.72] | 95 [74.0 to 99.87] | 19 [5.4 to 41.9] | 17 [3.6 to 41.4] | 24 [6.8 to 49.9]
  5/99 (Day 30, N=21,22,16,20,11,19,21,18,16) | 100 [83.9 to 100.0] | 86 [65.1 to 97.1] | 100 [79.4 to 100.0] | 90 [68.3 to 98.8] | 100 [71.5 to 100.0] | 100 [82.4 to 100.0] | 76 [52.8 to 91.8] | 83 [58.6 to 96.4] | 25 [7.3 to 52.4]
  5/99 (Day 365, N=21,22,16,20,11,19,21,18,17) | 95 [76.2 to 99.88] | 77 [54.6 to 92.2] | 100 [79.4 to 100.0] | 80 [56.3 to 94.3] | 100 [71.5 to 100.0] | 100 [82.4 to 100.0] | 43 [21.8 to 66.0] | 33 [13.3 to 59.0] | 18 [3.8 to 43.4]
  H44/76 (Day 1, N=21,22,15,20,11,20,21,18,17) | 19 [5.4 to 41.9] | 27 [10.7 to 50.2] | 13 [1.7 to 40.5] | 15 [3.2 to 37.9] | 45 [16.7 to 76.6] | 30 [11.9 to 54.3] | 5 [0.12 to 23.8] | 6 [0.14 to 27.3] | 0 [0.0 to 19.5]
  H44/76 (Day 30, N=21,22,16,20,11,20,19,18,16) | 95 [76.2 to 99.88] | 27 [10.7 to 50.2] | 100 [79.4 to 100.0] | 15 [3.2 to 37.9] | 100 [71.5 to 100.0] | 100 [83.2 to 100.0] | 58 [33.5 to 79.7] | 33 [13.3 to 59.0] | 6 [0.16 to 30.2]
  H44/76 (Day 365, N=21,22,16,20,11,20,21,18,17) | 76 [52.8 to 91.8] | 18 [5.2 to 40.3] | 44 [19.8 to 70.1] | 10 [1.2 to 31.7] | 82 [48.2 to 97.7] | 65 [40.8 to 84.6] | 19 [5.4 to 41.9] | 11 [1.4 to 34.7] | 6 [0.15 to 28.7]
  M01-0240364 (Day 1, N=21,22,14,18,10,19,20,17,17) | 24 [8.2 to 47.2] | 27 [10.7 to 50.2] | 21 [4.7 to 50.8] | 6 [0.14 to 27.3] | 20 [2.5 to 55.6] | 42 [20.3 to 66.5] | 5 [0.13 to 24.9] | 6 [0.15 to 28.7] | 12 [1.5 to 36.4]
  M01-0240364 (Day 30, N=21,22,16,17,11,19,19,18,16) | 100 [83.9 to 100.0] | 27 [10.7 to 50.2] | 100 [79.4 to 100.0] | 6 [0.15 to 28.7] | 100 [71.5 to 100.0] | 100 [82.4 to 100.0] | 21 [6.1 to 45.6] | 28 [9.7 to 53.5] | 13 [1.6 to 38.3]
  M01-0240364(Day 365, N=21,22,16,18,11,19,20,18,17) | 71 [47.8 to 88.7] | 32 [13.9 to 54.9] | 75 [47.6 to 92.7] | 6 [0.14 to 27.3] | 100 [71.5 to 100.0] | 95 [74.0 to 99.87] | 15 [3.2 to 37.9] | 11 [1.4 to 34.7] | 18 [3.8 to 43.4]
  M07-0241084 (Day 1, N=21,22,14,20,11,19,21,18,17) | 38 [18.1 to 61.6] | 41 [20.7 to 63.6] | 29 [8.4 to 58.1] | 25 [8.7 to 49.1] | 64 [30.8 to 89.1] | 58 [33.5 to 79.7] | 19 [5.4 to 41.9] | 17 [3.6 to 41.4] | 35 [14.2 to 61.7]
  M07-0241084 (Day 30, N=21,22,16,20,11,19,21,18,16) | 100 [83.9 to 100.0] | 45 [24.4 to 67.8] | 94 [69.8 to 99.84] | 25 [8.7 to 49.1] | 91 [58.7 to 99.77] | 95 [74.0 to 99.87] | 33 [14.6 to 57.0] | 22 [6.4 to 47.6] | 38 [15.2 to 64.6]
  M07-0241084(Day 365, N=21,22,16,20,11,19,21,18,17) | 62 [38.4 to 81.9] | 32 [13.9 to 54.9] | 50 [24.7 to 75.3] | 20 [5.7 to 43.7] | 82 [48.2 to 97.7] | 74 [48.8 to 90.9] | 29 [11.3 to 52.2] | 17 [3.6 to 41.4] | 35 [14.2 to 61.7]
  M14459 (Day 1, N=21,22,14,20,11,20,21,18,17) | 24 [8.2 to 47.2] | 36 [17.2 to 59.3] | 7 [0.18 to 33.9] | 15 [3.2 to 37.9] | 36 [10.9 to 69.2] | 30 [11.9 to 54.3] | 10 [1.2 to 30.4] | 11 [1.4 to 34.7] | 24 [6.8 to 49.9]
  M14459 (Day 30, N=21,22,16,20,11,20,20,18,16) | 95 [76.2 to 99.88] | 32 [13.9 to 54.9] | 88 [61.7 to 98.4] | 20 [5.7 to 43.7] | 100 [71.5 to 100.0] | 95 [75.1 to 99.87] | 35 [15.4 to 59.2] | 33 [13.3 to 59.0] | 25 [7.3 to 52.4]
  M14459 (Day 365, N=21,22,16,20,11,20,21,18,17) | 57 [34.0 to 78.2] | 18 [5.2 to 40.3] | 38 [15.2 to 64.6] | 5 [0.13 to 24.9] | 82 [48.2 to 97.7] | 60 [36.1 to 80.9] | 14 [3.0 to 36.3] | 11 [1.4 to 34.7] | 24 [6.8 to 49.9]
  NZ98/254 (Day 1, N=21,22,14,20,11,19,21,18,17) | 19 [5.4 to 41.9] | 32 [13.9 to 54.9] | 7 [0.18 to 33.9] | 5 [0.13 to 24.9] | 9 [0.23 to 41.3] | 26 [9.1 to 51.2] | 5 [0.12 to 23.8] | 6 [0.14 to 27.3] | 0 [0.0 to 19.5]
  NZ98/254 (Day 30, N=21,22,16,20,11,19,21,18,16) | 95 [76.2 to 99.88] | 23 [7.8 to 45.4] | 75 [47.6 to 92.7] | 10 [1.2 to 31.7] | 82 [48.2 to 97.7] | 95 [74.0 to 99.87] | 19 [5.4 to 41.9] | 17 [3.6 to 41.4] | 6 [0.16 to 30.2]
  NZ98/254 (Day 365, N=21,22,16,20,11,19,21,18,17) | 29 [11.3 to 52.2] | 14 [2.9 to 34.9] | 31 [11.0 to 58.7] | 5 [0.13 to 24.9] | 45 [16.7 to 76.6] | 42 [20.3 to 66.5] | 19 [5.4 to 41.9] | 6 [0.14 to 27.3] | 6 [0.15 to 28.7]

15. Secondary Outcome: 15. Percentage of Subjects With Four-fold Rise in HT-hSBA Titers Against N. Meningitidis Serogroup B Strains.
Description: Percentage of subjects with four-fold rise in HT-hSBA titers against N. meningitidis serogroup B strains, at 24 and 36 months after the primary vaccination.
  Four-fold rise is defined as follows: for subjects with a pre-vaccination titer < 1:2, a post-titer of ≥ 1:8; for subjects with a pre-vaccination titer ≥ 1:2 at least a four-fold increase.
Time Frame: Day 1, Day 30 and Day 365
Population: Analysis was done on FAS Day 365 (Persistence of Booster). All subjects in the enrolled population who were randomized, actually received the study vaccination in V102_03E1 and provided an evaluable serum sample at Day 365.
Measure: Number (95% Confidence Interval); unit: Percentages of Subjects
Arm/Group | 2OMV_OMV | 2OMV_Pbo | 2qOMV_qOMV | 2qOMV_Pbo | 2B_OMV | 2B_qOMV | 1M_OMV | 1M_qOMV | 1M_Pbo
Number analyzed (Participants) | 21 | 22 | 15 | 20 | 11 | 19 | 21 | 18 | 17
Percentages of Subjects
  5/99 (Day 1, N= 20,21,15,19,11,18,6,4,5) | 95 [75.1 to 99.87] | 100 [83.9 to 100.0] | 100 [78.2 to 100.0] | 100 [82.4 to 100.0] | 91 [58.7 to 99.77] | 94 [72.7 to 99.86] | 0 [0.0 to 45.9] | 0 [0.0 to 60.2] | 0 [0.0 to 52.2]
  5/99 (Day 30, N=21,22,14,20,9,19,21,18,16) | 100 [83.9 to 100.0] | 5 [0.12 to 22.8] | 93 [66.1 to 99.82] | 0 [0.0 to 16.8] | 100 [66.4 to 100.0] | 100 [82.4 to 100.0] | 57 [34.0 to 78.2] | 78 [52.4 to 93.6] | 6 [0.16 to 30.2]
  5/99 (Day 365, N=21,22,14,20,9,19,21,18,17) | 67 [43.0 to 85.4] | 5 [0.12 to 22.8] | 86 [57.2 to 98.2] | 0 [0.0 to 16.8] | 89 [51.8 to 99.72] | 74 [48.8 to 90.9] | 29 [11.3 to 52.2] | 28 [9.7 to 53.5] | 6 [0.15 to 28.7]
  H44/76 (Day 1, N=20,22,15,20,11,19,6,4,5) | 100 [83.2 to 100.0] | 95 [77.2 to 99.88] | 100 [78.2 to 100.0] | 95 [75.1 to 99.87] | 91 [58.7 to 99.77] | 89 [66.9 to 98.7] | 0 [0.0 to 45.9] | 0 [0.0 to 60.2] | 0 [0.0 to 52.2]
  H44/76 (Day 30, N=21,22,15,20,11,20,19,18,16) | 81 [58.1 to 94.6] | 5 [0.12 to 22.8] | 93 [68.1 to 99.83] | 0 [0.0 to 16.8] | 100 [71.5 to 100.0] | 75 [50.9 to 91.3] | 37 [16.3 to 61.6] | 28 [9.7 to 53.5] | 6 [0.16 to 30.2]
  H44/76 (Day 365, N=21,22,15,20,11,20,21,18,17) | 38 [18.1 to 61.6] | 0 [0.0 to 15.4] | 20 [4.3 to 48.1] | 0 [0.0 to 16.8] | 64 [30.8 to 89.1] | 30 [11.9 to 54.3] | 10 [1.2 to 30.4] | 0 [0.0 to 18.5] | 6 [0.15 to 28.7]
  M01-0240364 (Day 1, N=19,21,15,15,11,18,6,4,4) | 79 [54.4 to 93.9] | 76 [52.8 to 91.8] | 67 [38.4 to 88.2] | 67 [38.4 to 88.2] | 82 [48.2 to 97.7] | 89 [65.3 to 98.6] | 0 [0.0 to 45.9] | 0 [0.0 to 60.2] | 0 [0.0 to 60.2]
  M01-0240364 (Day 30, N=21,22,14,17,10,19,19,17,16) | 100 [83.9 to 100.0] | 5 [0.12 to 22.8] | 93 [66.1 to 99.82] | 6 [0.15 to 28.7] | 100 [69.2 to 100.0] | 89 [66.9 to 98.7] | 16 [3.4 to 39.6] | 24 [6.8 to 49.9] | 6 [0.16 to 30.2]
  M01-0240364 (Day 365,N=21,22,14,18,10,19,20,17,17) | 62 [38.4 to 81.9] | 5 [0.12 to 22.8] | 64 [35.1 to 87.2] | 6 [0.14 to 27.3] | 90 [55.5 to 99.75] | 79 [54.4 to 93.9] | 15 [3.2 to 37.9] | 6 [0.15 to 28.7] | 6 [0.15 to 28.7]
  M07-0241084 (Day 1, N=20,20,15,18,11,18,6,4,4) | 30 [11.9 to 54.3] | 20 [5.7 to 43.7] | 33 [11.8 to 61.6] | 17 [3.6 to 41.4] | 45 [16.7 to 76.6] | 56 [30.8 to 78.5] | 0 [0.0 to 45.9] | 0 [0.0 to 60.2] | 0 [0.0 to 60.2]
  M07-0241084 (Day 30, N=21,22,14,20,11,19,21,18,16) | 81 [58.1 to 94.6] | 0 [0.0 to 15.4] | 93 [66.1 to 99.82] | 0 [0.0 to 16.8] | 82 [48.2 to 97.7] | 58 [33.5 to 79.7] | 14 [3.0 to 36.3] | 0 [0.0 to 18.5] | 6 [0.16 to 30.2]
  M07-0241084 (Day 365,N=21,22,14,20,11,19,21,18,17) | 19 [5.4 to 41.9] | 0 [0.0 to 15.4] | 0 [0.0 to 23.2] | 0 [0.0 to 16.8] | 27 [6.0 to 61.0] | 5 [0.13 to 26.0] | 0 [0.0 to 16.1] | 0 [0.0 to 18.5] | 6 [0.15 to 28.7]
  M14459 (Day 1, N=20,22,15,19,11,19,6,4,5) | 55 [31.5 to 76.9] | 55 [32.2 to 75.6] | 67 [38.4 to 88.2] | 58 [33.5 to 79.7] | 91 [58.7 to 99.77] | 63 [38.4 to 83.7] | 0 [0.0 to 45.9] | 0 [0.0 to 60.2] | 0 [0.0 to 52.2]
  M14459 (Day 30, N=21,22,14,20,11,20,20,18,16) | 76 [52.8 to 91.8] | 0 [0.0 to 15.4] | 86 [57.2 to 98.2] | 0 [0.0 to 16.8] | 100 [71.5 to 100.0] | 75 [50.9 to 91.3] | 15 [3.2 to 37.9] | 6 [0.14 to 27.3] | 6 [0.16 to 30.2]
  M14459 (Day 365, N=21,22,14,20,11,20,21,18,17) | 24 [8.2 to 47.2] | 0 [0.0 to 15.4] | 0 [0.0 to 23.2] | 0 [0.0 to 16.8] | 36 [10.9 to 69.2] | 25 [8.7 to 49.1] | 10 [1.2 to 30.4] | 0 [0.0 to 18.5] | 6 [0.15 to 28.7]
  NZ98/254 (Day 1, N=20,21,15,19,11,18,6,4,5) | 60 [36.1 to 80.9] | 52 [29.8 to 74.3] | 53 [26.6 to 78.7] | 58 [33.5 to 79.7] | 55 [23.4 to 83.3] | 67 [41.0 to 86.7] | 0 [0.0 to 45.9] | 0 [0.0 to 60.2] | 0 [0.0 to 52.2]
  NZ98/254 (Day 30, N=21,22,14,20,11,19,21,18,16) | 81 [58.1 to 94.6] | 0 [0.0 to 15.4] | 71 [41.9 to 91.6] | 5 [0.13 to 24.9] | 82 [48.2 to 97.7] | 63 [38.4 to 83.7] | 19 [5.4 to 41.9] | 6 [0.14 to 27.3] | 6 [0.16 to 30.2]
  NZ98/254 (Day 365, N=21,22,14,20,11,19,21,18,17) | 10 [1.2 to 30.4] | 0 [0.0 to 15.4] | 14 [1.8 to 42.8] | 0 [0.0 to 16.8] | 9 [0.23 to 41.3] | 5 [0.13 to 26.0] | 10 [1.2 to 30.4] | 0 [0.0 to 18.5] | 6 [0.15 to 28.7]

16. Secondary Outcome: 16. The HT-hSBA GMTs Against N. Meningitidis Serogroups A, C, W, Y.
Description: The HT-hSBA GMTs against N. meningitidis serogroup A, C, W, Y, at 24 and 36 months after the primary vaccination.
Time Frame: Day 1 and Day 365
Population: as for outcome 15
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | 2OMV_OMV | 2OMV_Pbo | 2qOMV_qOMV | 2qOMV_Pbo | 2B_OMV | 2B_qOMV | 1M_OMV | 1M_qOMV | 1M_Pbo
Number analyzed (Participants) | 21 | 22 | 16 | 20 | 11 | 20 | 20 | 18 | 17
Titers
  Men A (Day 1, N=21,22,15,20,10,20,20,17,17) | 3.98 [1.98 to 8] | 2.73 [1.44 to 5.15] | 3.07 [1.26 to 7.47] | 2.98 [1.38 to 6.42] | 2.27 [0.87 to 5.94] | 4.22 [1.63 to 11] | 6.31 [2.82 to 14] | 2.49 [1.52 to 4.09] | 5.48 [2.18 to 14]
  Men A (Day 365, N=21,22,16,20,10,20,20,18,17) | 25 [11 to 59] | 2.62 [1.39 to 4.94] | 44 [18 to 105] | 3.03 [1.30 to 7.06] | 54 [17 to 174] | 53 [22 to 130] | 34 [16 to 69] | 6.52 [2.71 to 16] | 3.54 [1.40 to 8.92]
  Men C (Day 1, N=20,19,14,20,11,19,19,18,16) | 18 [8.21 to 39] | 19 [7.54 to 49] | 19 [8.13 to 44] | 10 [5.52 to 19] | 5.20 [2.80 to 9.65] | 7.83 [4.51 to 14] | 7.89 [4.26 to 15] | 8.45 [2.64 to 27] | 24 [9.34 to 61]
  Men C (Day 365, N=21,21,16,20,11,19,19,18,17) | 128 [75 to 217] | 15 [5.82 to 39] | 177 [102 to 305] | 9.14 [4.07 to 21] | 29 [10 to 82] | 32 [16 to 67] | 81 [46 to 141] | 72 [27 to 191] | 24 [8.98 to 66]
  Men W (Day 1, N=20,22,12,20,11,20,17,18,16) | 36 [21 to 62] | 43 [24 to 79] | 30 [7.82 to 112] | 17 [6.88 to 43] | 25 [7.98 to 79] | 23 [9.81 to 52] | 28 [11 to 70] | 15 [4.54 to 47] | 10 [3.53 to 30]
  Men W (Day 365, N=21,22,16,20,11,20,19,18,17) | 190 [133 to 272] | 28 [13 to 59] | 213 [135 to 337] | 16 [5.58 to 47] | 80 [26 to 246] | 96 [72 to 127] | 172 [97 to 306] | 104 [49 to 221] | 16 [5.27 to 49]
  Men Y (Day 1, N=21,21,14,20,11,18,20,18,17) | 10 [4.39 to 24] | 16 [4.85 to 54] | 24 [6.62 to 90] | 5.39 [2.06 to 14] | 2.40 [1.05 to 5.47] | 1.90 [1.02 to 3.55] | 7.05 [3.08 to 16] | 6.83 [2.11 to 22] | 7.03 [1.99 to 25]
  Men Y (Day 365, N=21,21,16,20,11,18,20,18,17) | 116 [58 to 231] | 18 [5.05 to 62] | 235 [147 to 376] | 5.93 [1.97 to 18] | 7.17 [1.91 to 27] | 20 [6.92 to 58] | 193 [123 to 301] | 101 [36 to 280] | 9.56 [2.44 to 37]

17. Secondary Outcome: 17. The HT-hSBA GMTs Against N. Meningitidis Strains of Serogroups B.
Description: The HT-hSBA GMTs against N. meningitidis strains of serogroups B, at 24 and 36 months after the primary vaccination.
Time Frame: Day 1 and Day 365
Population: as for outcome 14
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | 2OMV_OMV | 2OMV_Pbo | 2qOMV_qOMV | 2qOMV_Pbo | 2B_OMV | 2B_qOMV | 1M_OMV | 1M_qOMV | 1M_Pbo
Number analyzed (Participants) | 21 | 22 | 16 | 20 | 11 | 20 | 21 | 18 | 17
Titers
  5/99 (Day 1, N= 21,22,14,20,9,19,21,18,17) | 18 [9.47 to 34] | 18 [9.50 to 34] | 31 [12 to 85] | 31 [15 to 65] | 27 [8.61 to 86] | 39 [21 to 74] | 2.97 [1.58 to 5.59] | 1.80 [1.01 to 3.22] | 3.20 [1.44 to 7.09]
  5/99 (Day 365, N= 21,22,16,20,11,19,21,18,17) | 175 [79 to 385] | 13 [6.07 to 29] | 305 [149 to 625] | 23 [11 to 47] | 587 [351 to 983] | 491 [258 to 936] | 6.05 [3.10 to 12] | 4.23 [1.48 to 12] | 2.45 [1 to 5.99]
  H44/76 (Day 1, N= 21,22,15,20,11,20,21,18,17) | 3.58 [1.66 to 7.71] | 2.23 [1.28 to 3.90] | 1.49 [0.96 to 2.33] | 1.73 [0.97 to 3.10] | 3.45 [1.81 to 6.57] | 3.43 [1.83 to 6.43] | 1.34 [0.85 to 2.13] | 1.51 [0.91 to 2.48] | 1.19 [0.97 to 1.47]
  H44/76 (Day 365, N= 21,22,16,20,11,20,21,18,17) | 12 [5.18 to 26] | 1.93 [1.20 to 3.10] | 4.19 [1.93 to 9.11] | 1.83 [1.07 to 3.15] | 21 [6.00 to 71] | 11 [4.68 to 25] | 1.96 [1.21 to 3.19] | 1.92 [1.17 to 3.17] | 1.49 [0.90 to 2.48]
  M01-0240364 (Day 1, N= 21,22,14,18,10,19,20,17,17) | 2.33 [1.25 to 4.36] | 3.39 [1.43 to 8.05] | 2.87 [0.86 to 9.59] | 1.26 [0.89 to 1.80] | 2.46 [0.72 to 8.40] | 6.29 [2.22 to 18] | 1.24 [0.79 to 1.94] | 1.24 [0.88 to 1.77] | 1.68 [0.85 to 3.33]
  M01-0240364(Day 365,N= 21,22,16,18,11,19,20,18,17) | 30 [9.54 to 93] | 3.55 [1.56 to 8.07] | 74 [18 to 300] | 1.23 [0.91 to 1.68] | 303 [174 to 527] | 155 [69 to 350] | 1.61 [0.99 to 2.63] | 1.71 [0.86 to 3.42] | 2.03 [0.90 to 4.58]
  M07-0241084 (Day 1, N= 21,22,14,20,11,19,21,18,17) | 3.68 [2.07 to 6.54] | 4.20 [2.25 to 7.85] | 2.28 [1.16 to 4.48] | 2.36 [1.51 to 3.70] | 4.10 [1.89 to 8.90] | 7.35 [3.82 to 14] | 2.08 [1.26 to 3.42] | 2.15 [1.14 to 4.05] | 3.50 [1.57 to 7.80]
  M07-0241084 (Day 365,N=21,22,16,20,11,19,21,18,17) | 7.96 [4.60 to 14] | 3.28 [2.16 to 4.97] | 4.09 [2.30 to 7.25] | 2.04 [1.43 to 2.92] | 10 [4.51 to 24] | 11 [6.35 to 18] | 2.45 [1.59 to 3.79] | 1.91 [1.14 to 3.23] | 3.92 [1.90 to 8.07]
  M14459 (Day 1, N= 21,22,14,20,11,20,21,18,16) | 2.69 [1.51 to 4.78] | 2.94 [1.77 to 4.89] | 1.54 [0.90 to 2.63] | 2.01 [1.40 to 2.88] | 3.11 [1.74 to 5.56] | 3.37 [1.95 to 5.81] | 1.85 [1.13 to 3.04] | 1.48 [1.03 to 2.13] | 2.55 [1.37 to 4.77]
  M14459 (Day 365, N= 21,22,16,20,11,20,21,18,17) | 7.19 [3.89 to 13] | 1.67 [1.07 to 2.60] | 2.94 [1.49 to 5.80] | 1.47 [1.07 to 2.03] | 11 [4.41 to 28] | 7.12 [3.59 to 14] | 2.09 [1.33 to 3.29] | 1.38 [0.98 to 1.93] | 2.17 [1.07 to 4.41]
  NZ98/254 (Day 1, N= 21,22,14,20,11,19,21,18,17) | 1.73 [1.06 to 2.81] | 2.34 [1.33 to 4.10] | 1.34 [0.94 to 1.93] | 1.48 [1.01 to 2.17] | 1.72 [0.99 to 2.98] | 2.24 [1.20 to 4.17] | 1.18 [0.84 to 1.66] | 1.19 [0.90 to 1.58] | 1.13 [0.94 to 1.37]
  NZ98/254 (Day 365, N= 21,22,16,20,11,19,21,18,17) | 3.49 [2.12 to 5.74] | 1.71 [1.41 to 2.57] | 2.67 [1.27 to 5.61] | 1.23 [0.90 to 1.69] | 3.28 [1.66 to 6.49] | 3.77 [1.98 to 7.18] | 1.65 [1.04 to 2.61] | 1.19 [0.91 to 1.54] | 1.28 [0.85 to 1.92]

18. Secondary Outcome: 18. Percentage of Subjects With HT-hSBA Titer ≥ 1:8 to N. Meningitidis Serogroups A, C, W,Y.
Description: Percentage of subjects with HT-hSBA titer ≥ 1:8 against N. meningitidis serogroups A, C, W, Y at Day 1, Day 30 (one month) and Day 365 (12 months) after the administration of MenABCWY booster vaccination.
Time Frame: Day 1, Day 30 and Day 365
Population: as for outcome 15
Measure: Number (95% Confidence Interval); unit: Percentages of Subjects
Arm/Group | 2OMV_OMV | 2OMV_Pbo | 2qOMV_qOMV | 2qOMV_Pbo | 2B_OMV | 2B_qOMV | 1M_OMV | 1M_qOMV | 1M_Pbo
Number analyzed (Participants) | 21 | 22 | 16 | 20 | 11 | 20 | 20 | 18 | 17
Percentages of Subjects
  Men A (Day 1,N=21,22,15,20,10,20,20,17,17) | 38 [18.1 to 61.6] | 18 [5.2 to 40.3] | 20 [4.3 to 48.1] | 30 [11.9 to 54.3] | 30 [6.7 to 65.2] | 35 [15.4 to 59.2] | 45 [23.1 to 68.5] | 12 [1.5 to 36.4] | 41 [18.4 to 67.1]
  Men A (Day 30, N=21,22,15,19,10,20,18,16,16) | 100 [83.9 to 100.0] | 32 [13.9 to 54.9] | 100 [78.2 to 100.0] | 26 [9.1 to 51.2] | 100 [69.2 to 100.0] | 95 [75.1 to 99.87] | 100 [81.5 to 100.0] | 94 [69.8 to 99.84] | 44 [19.8 to 70.1]
  Men A (Day 365, N=21,22,16,20,10,20,20,18,17) | 67 [43.0 to 85.4] | 23 [7.8 to 45.4] | 88 [61.7 to 98.4] | 25 [8.7 to 49.1] | 90 [55.5 to 99.75] | 85 [62.1 to 96.8] | 85 [62.1 to 96.8] | 50 [26.0 to 74.0] | 35 [14.2 to 61.7]
  Men C (Day 1, N=20,19,14,20,11,19,19,18,16) | 65 [40.8 to 84.6] | 68 [43.4 to 87.4] | 71 [41.9 to 91.6] | 65 [40.8 to 84.6] | 36 [10.9 to 69.2] | 58 [33.5 to 79.7] | 58 [33.5 to 79.7] | 50 [26.0 to 74.0] | 75 [47.6 to 92.7]
  Men C (Day 30, N=17,20,10,20,7,14,19,17,16) | 100 [80.5 to 100.0] | 65 [40.8 to 84.6] | 100 [69.2 to 100.0] | 55 [31.5 to 76.9] | 100 [59.0 to 100.0] | 100 [76.8 to 100.0] | 100 [82.4 to 100.0] | 88 [63.6 to 98.5] | 69 [41.3 to 89.0]
  Men C (Day 365, N=21,21,16,20,11,19,19,18,17) | 100 [83.9 to 100.0] | 62 [38.4 to 81.9] | 100 [79.4 to 100.0] | 50 [27.2 to 72.8] | 82 [48.2 to 97.7] | 95 [74.0 to 99.87] | 100 [82.4 to 100.0] | 89 [65.3 to 98.6] | 65 [38.3 to 85.8]
  Men W (Day 1,N=20,22,12,20,11,20,17,18,16) | 95 [75.1 to 99.87] | 95 [77.2 to 99.88] | 75 [42.8 to 94.5] | 70 [45.7 to 88.1] | 82 [48.2 to 97.7] | 75 [50.9 to 91.3] | 82 [56.6 to 96.2] | 61 [35.7 to 82.7] | 56 [29.9 to 80.2]
  Men W (Day 30, N=18,22,15,19,11,18,17,16,14) | 100 [81.5 to 100.0] | 86 [65.1 to 97.1] | 100 [78.2 to 100.0] | 74 [48.8 to 90.9] | 100 [71.5 to 100.0] | 100 [81.5 to 100.0] | 100 [80.5 to 100.0] | 100 [79.4 to 100.0] | 57 [28.9 to 82.3]
  Men W (Day 365, N=21,22,16,20,11,20,19,18,17) | 100 [83.9 to 100.0] | 82 [59.7 to 94.8] | 100 [79.4 to 100.0] | 65 [40.8 to 84.6] | 91 [58.7 to 99.77] | 100 [83.2 to 100.0] | 100 [82.4 to 100.0] | 100 [81.5 to 100.0] | 65 [38.3 to 85.8]
  Men Y (Day 1, N=21,21,14,20,11,18,20,18,17) | 62 [38.4 to 81.9] | 62 [38.4 to 81.9] | 71 [41.9 to 91.6] | 40 [19.1 to 63.9] | 36 [10.9 to 69.2] | 11 [1.4 to 34.7] | 55 [31.5 to 76.9] | 44 [21.5 to 69.2] | 41 [18.4 to 67.1]
  Men Y (Day 30, N=21,21,15,20,11,18,20,17,16) | 100 [83.9 to 100.0] | 57 [34.0 to 78.2] | 100 [78.2 to 100.0] | 40 [19.1 to 63.9] | 82 [48.2 to 97.7] | 83 [58.6 to 96.4] | 100 [83.2 to 100.0] | 100 [80.5 to 100.0] | 38 [15.2 to 64.6]
  Men Y (Day 365, N=21,21,16,20,11,18,20,18,17) | 95 [76.2 to 99.88] | 52 [29.8 to 74.3] | 100 [79.4 to 100.0] | 40 [19.1 to 63.9] | 45 [16.7 to 76.6] | 72 [46.5 to 90.3] | 100 [83.2 to 100.0] | 89 [65.3 to 98.6] | 47 [23.0 to 72.2]

19. Secondary Outcome: 19. Percentage of Subjects With HT-hSBA Titer ≥ 1:5 to N. Meningitidis Strains of Serogroup B.
Description: Percentage of subjects with HT-hSBA titer ≥ 1:5 against N. meningitides strains of serogroups B at Day 1, Day 30 (one month) and Day 365 (12 months) after the administration of MenABCWY booster vaccination.
Time Frame: Day 1, Day 30 and Day 365
Population: as for outcome 15
Measure: Number (95% Confidence Interval); unit: Percentages of Subjects
Arm/Group | 2OMV_OMV | 2qOMV_qOMV | 2B_OMV | 2B_qOMV | 1M_OMV | 1M_qOMV
Number analyzed (Participants) | 21 | 16 | 11 | 20 | 21 | 18
Percentages of Subjects
  5/99 (Day 1,N= 21,14,9,19,21,18) | 76 [52.8 to 91.8] | 86 [57.2 to 98.2] | 89 [51.8 to 99.72] | 95 [74 to 99.87] | 19 [5.4 to 41.9] | 17 [3.6 to 41.4]
  5/99 (Day 30, N= 21,16,11,19,21,18) | 100 [83.9 to 100] | 100 [79.4 to 100] | 100 [71.5 to 100] | 100 [82.4 to 100] | 76 [52.8 to 91.8] | 83 [58.6 to 96.4]
  5/99 (Day 365, 21,16,11,19,21,18) | 95 [76.2 to 99.88] | 100 [79.4 to 100] | 100 [71.5 to 100] | 100 [82.4 to 100] | 43 [21.8 to 66] | 33 [13.3 to 59]
  H44/76 (Day 1, N= 21,15,11,20,21,18) | 19 [5.4 to 41.9] | 13 [1.7 to 40.5] | 45 [16.7 to 76.6] | 30 [11.9 to 54.3] | 5 [0.12 to 23.8] | 6 [0.14 to 27.3]
  H44/76 (Day 30, N= 21,16,11,20,19,18) | 95 [76.2 to 99.88] | 100 [79.4 to 100] | 100 [71.5 to 100] | 100 [83.2 to 100] | 58 [33.5 to 79.7] | 33 [13.3 to 59]
  H44/76 (Day 365, N= 21,16,11,20,21,18) | 76 [52.8 to 91.8] | 44 [19.8 to 70.1] | 82 [48.2 to 97.7] | 65 [40.8 to 84.6] | 19 [5.4 to 41.9] | 11 [1.4 to 34.7]
  M01-0240364 (Day 1, N= 21,14,10,19,20,17) | 24 [8.2 to 47.2] | 21 [4.7 to 50.8] | 20 [2.5 to 55.6] | 42 [20.3 to 66.5] | 5 [0.13 to 24.9] | 6 [0.15 to 28.7]
  M01-0240364(Day 30, N= 21,16,11,19,19,18) | 100 [83.9 to 100] | 100 [79.4 to 100] | 100 [71.5 to 100] | 100 [82.4 to 100] | 21 [6.1 to 45.6] | 28 [9.7 to 53.5]
  M01-0240364 (Day 365, N= 21,16,11,19,20,18) | 71 [47.8 to 88.7] | 75 [47.6 to 92.7] | 100 [71.5 to 100] | 95 [74 to 99.87] | 15 [3.2 to 37.9] | 11 [1.4 to 34.7]
  M07-0241084 (Day 1, N= 21,14,11,19,21,18) | 38 [18.1 to 61.6] | 29 [8.4 to 58.1] | 64 [30.8 to 89.1] | 58 [33.5 to 79.7] | 19 [5.4 to 41.9] | 17 [3.6 to 41.4]
  M07-0241084 (Day 30, N= 21,16,11,19,21,18) | 100 [83.9 to 100] | 94 [69.8 to 99.84] | 91 [58.7 to 99.77] | 95 [74 to 99.87] | 33 [14.6 to 57] | 22 [6.4 to 47.6]
  M07-0241084(Day 365, N=21,16,11,19,21,18) | 62 [38.4 to 81.9] | 50 [24.7 to 75.3] | 82 [48.2 to 97.7] | 74 [48.8 to 90.9] | 29 [11.3 to 52.2] | 17 [3.6 to 41.4]
  M14459 (Day 1, N= 21,14,11,20,21,18) | 24 [8.2 to 47.2] | 7 [0.18 to 33.9] | 36 [10.9 to 69.2] | 30 [11.9 to 54.3] | 10 [1.2 to 30.4] | 11 [1.4 to 34.7]
  M14459 (Day 30, N= 21,16,11,20,20,18) | 95 [76.2 to 99.88] | 88 [61.7 to 98.4] | 100 [71.5 to 100] | 95 [75.1 to 99.87] | 35 [15.4 to 59.2] | 33 [13.3 to 59]
  M14459 (Day 365, N= 21,16,11,20,21,18) | 57 [34 to 78.2] | 38 [15.2 to 64.6] | 82 [48.2 to 97.7] | 60 [36.1 to 80.9] | 14 [3 to 36.3] | 11 [1.4 to 34.7]
  NZ98/254 (Day 1,N= 21,14,11,19,21,18) | 19 [5.4 to 41.9] | 7 [0.18 to 33.9] | 9 [0.23 to 41.3] | 26 [9.1 to 51.2] | 5 [0.12 to 23.8] | 6 [0.14 to 27.3]
  NZ98/254 (Day 30, N= 21,16,11,19,21,18) | 95 [76.2 to 99.88] | 75 [47.6 to 92.7] | 82 [48.2 to 97.7] | 95 [74 to 99.87] | 19 [5.4 to 41.9] | 17 [3.6 to 41.4]
  NZ98/254 (Day 365, N= 21,16,11,19,21,18) | 29 [11.3 to 52.2] | 31 [11 to 58.7] | 45 [16.7 to 76.6] | 42 [20.3 to 66.5] | 19 [5.4 to 41.9] | 6 [0.14 to 27.3]

20. Secondary Outcome: 20. The HT-hSBA GMTs Against Neisseria Meningitidis Serogroups A, C, W,Y and Strains of Serogroups B.
Description: The HT-hSBA GMTs against Neisseria meningitidis serogroup A, C, W, Y and strains of serogroups B at Day 1, Day 30 (one month) and Day 365 (12 months) after the administration of MenABCWY booster vaccination.
Time Frame: Day 1, Day 30 and Day 365
Population: as for outcome 15
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | 2OMV_OMV | 2OMV_Pbo | 2qOMV_qOMV | 2qOMV_Pbo | 2B_OMV | 2B_qOMV | 1M_OMV | 1M_qOMV | 1M_Pbo
Number analyzed (Participants) | 21 | 22 | 16 | 20 | 11 | 20 | 20 | 18 | 17
Titers
  Men A (Day 1, N= 21,22,15,20,10,20,20,17,17) | 3.98 [1.98 to 8] | 2.73 [1.44 to 5.15] | 3.07 [1.26 to 7.47] | 2.98 [1.38 to 6.42] | 2.27 [0.87 to 5.94] | 4.22 [1.63 to 11] | 6.31 [2.82 to 14] | 2.49 [1.52 to 4.09] | 5.48 [2.18 to 14]
  Men A (Day 30, N= 21,22,15,19,10,20,18,16,16) | 275 [174 to 435] | 3.88 [1.74 to 8.66] | 348 [202 to 601] | 2.95 [1.41 to 6.17] | 445 [277 to 715] | 428 [196 to 931] | 140 [82 to 239] | 46 [23 to 91] | 5.99 [2.27 to 16]
  Men A (Day 365, N= 21,22,16,20,10,20,20,18,17) | 25 [11 to 59] | 2.62 [1.39 to 4.94] | 44 [18 to 105] | 3.03 [1.30 to 7.06] | 54 [17 to 174] | 53 [22 to 130] | 34 [16 to 69] | 6.52 [2.71 to 16] | 3.54 [1.40 to 8.92]
  Men C (Day 1, N= 20,19,14,20,11,19,19,18,16) | 18 [8.21 to 39] | 19 [7.54 to 49] | 19 [8.13 to 44] | 10 [5.52 to 19] | 5.20 [2.80 to 9.65] | 7.83 [4.51 to 14] | 7.89 [4.26 to 15] | 8.45 [2.64 to 27] | 24 [9.34 to 61]
  Men C (Day 30, N= 17,20,10,20,7,14,19,17,16) | 737 [459 to 1183] | 21 [8.38 to 52] | 766 [325 to 1804] | 8.43 [4.37 to 16] | 292 [75 to 1142] | 102 [57 to 181] | 322 [186 to 556] | 307 [118 to 795] | 27 [9.15 to 78]
  Men C (Day 365, N= 21,21,16,20,11,19,19,18,17) | 128 [75 to 217] | 15 [5.82 to 39] | 177 [102 to 305] | 9.14 [4.07 to 21] | 29 [10 to 82] | 32 [16 to 67] | 81 [46 to 141] | 72 [27 to 191] | 24 [8.98 to 66]
  Men W (Day 1, N= 20,22,12,20,11,20,17,18,16) | 36 [21 to 62] | 43 [24 to 79] | 30 [7.82 to 112] | 17 [6.88 to 43] | 25 [7.98 to 79] | 23 [9.81 to 52] | 28 [11 to 70] | 15 [4.54 to 47] | 10 [3.53 to 30]
  Men W (Day 30, N= 18,22,15,19,11,18,17,16,14) | 844 [535 to 1333] | 46 [23 to 89] | 890 [665 to 1190] | 22 [8.89 to 52] | 392 [252 to 610] | 395 [321 to 487] | 620 [354 to 1085] | 360 [169 to 765] | 13 [3.50 to 52]
  Men W (Day 365, N= 21,22,16,20,11,20,19,18,17) | 190 [133 to 272] | 28 [13 to 59] | 213 [135 to 337] | 16 [5.58 to 47] | 80 [26 to 246] | 96 [72 to 127] | 172 [97 to 306] | 104 [49 to 221] | 16 [5.27 to 49]
  Men Y (Day 1, N= 21,21,14,20,11,18,20,18,17) | 10 [4.39 to 24] | 16 [4.85 to 54] | 24 [6.62 to 90] | 5.39 [2.06 to 14] | 2.40 [1.05 to 5.47] | 1.90 [1.02 to 3.55] | 7.05 [3.08 to 16] | 6.83 [2.11 to 22] | 7.03 [1.99 to 25]
  Men Y (Day 30, N= 21,21,15,20,11,18,20,17,16) | 444 [257 to 768] | 17 [4.77 to 57] | 748 [463 to 1208] | 4.86 [1.86 to 13] | 48 [14 to 157] | 54 [17 to 171] | 662 [424 to 1032] | 404 [201 to 811] | 6.84 [1.78 to 26]
  Men Y (Day 365, N= 21,21,16,20,11,18,20,18,17) | 116 [58 to 231] | 18 [5.05 to 62] | 235 [147 to 376] | 5.93 [1.97 to 18] | 7.17 [1.91 to 27] | 20 [6.92 to 58] | 193 [123 to 301] | 101 [36 to 280] | 9.56 [2.44 to 37]

21. Secondary Outcome: 21. The HT-hSBA GMTs Against Neisseria Meningitidis Strains of Serogroups B.
Description: The HT-hSBA GMTs against Neisseria meningitidis strains of serogroups B at Day 1, Day 30 (one month) and Day 365 (12 months) after the administration of MenABCWY booster vaccination.
Time Frame: Day 1, Day 30 and Day 365
Population: as for outcome 15
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | 2OMV_OMV | 2OMV_Pbo | 2qOMV_qOMV | 2qOMV_Pbo | 2B_OMV | 2B_qOMV | 1M_OMV | 1M_qOMV | 1M_Pbo
Number analyzed (Participants) | 21 | 22 | 16 | 20 | 11 | 20 | 21 | 18 | 17
Titers
  5/99 (Day 1, N=21,22,14,20,9,19,21,18,17) | 18 [9.47 to 34] | 18 [9.50 to 34] | 31 [12 to 85] | 31 [15 to 65] | 27 [8.61 to 86] | 39 [21 to 74] | 2.97 [1.58 to 5.59] | 1.8 [1.01 to 3.22] | 3.2 [1.44 to 7.09]
  5/99 (Day 30, N=21,22,16,20,11,19,21,18,16) | 1147 [665 to 1980] | 23 [11 to 48] | 1598 [864 to 2956] | 35 [19 to 65] | 2205 [1560 to 3117] | 2816 [1856 to 4273] | 28 [11 to 67] | 29 [10 to 80] | 3.98 [1.24 to 13]
  5/99 (Day 365, N=21,22,16,20,11,19,21,18,17) | 175 [79 to 385] | 13 [6.07 to 29] | 305 [149 to 625] | 23 [11 to 47] | 587 [351 to 983] | 491 [258 to 936] | 6.05 [3.10 to 12] | 4.23 [1.48 to 12] | 2.45 [1 to 5.99]
  H44/76 (Day 1, N=21,22,15,20,11,20,21,18,17) | 3.58 [1.66 to 7.71] | 2.23 [1.28 to 3.90] | 1.49 [0.96 to 2.33] | 1.73 [0.97 to 3.10] | 3.45 [1.81 to 6.57] | 3.43 [1.83 to 6.43] | 1.34 [0.85 to 2.13] | 1.51 [0.91 to 2.48] | 1.19 [0.97 to 1.47]
  H44/76 (Day 30, N=21,22,16,20,11,20,19,18,16) | 104 [59 to 184] | 2.65 [1.48 to 4.78] | 57 [32 to 102] | 2.03 [1.11 to 3.73] | 132 [64 to 271] | 79 [40 to 153] | 5.27 [2.54 to 11] | 3.89 [1.79 to 8.47] | 1.6 [0.67 to 3.83]
  H44/76 (Day 365, N=21,22,16,20,11,20,21,18,17) | 12 [5.18 to 26] | 1.93 [1.20 to 3.10] | 4.19 [1.93 to 9.11] | 1.83 [1.07 to 3.15] | 21 [6 to 71] | 11 [4.68 to 25] | 1.96 [1.21 to 3.19] | 1.92 [1.17 to 3.17] | 1.49 [0.90 to 2.48]
  M01-0240364 (Day 1, N=21,22,14,18,10,19,20,17,17) | 2.33 [1.25 to 4.36] | 3.39 [1.43 to 8.05] | 2.87 [0.86 to 9.59] | 1.26 [0.89 to 1.80] | 2.46 [0.72 to 8.40] | 6.29 [2.22 to 18] | 1.24 [0.79 to 1.94] | 1.24 [0.88 to 1.77] | 1.68 [0.85 to 3.33]
  M01-0240364 (Day 30, N=21,22,16,17,11,19,19,18,16) | 679 [352 to 1310] | 3.57 [1.39 to 9.14] | 903 [463 to 1761] | 1.23 [0.89 to 1.70] | 1336 [810 to 2202] | 1261 [746 to 2131] | 2.68 [1.15 to 6.25] | 3.66 [1.21 to 11] | 1.89 [0.72 to 4.91]
  M01-0240364 (Day 365,N=21,22,16,18,11,19,20,18,17) | 30 [9.54 to 93] | 3.55 [1.56 to 8.07] | 74 [18 to 300] | 1.23 [0.91 to 1.68] | 303 [174 to 527] | 155 [69 to 350] | 1.61 [0.99 to 2.63] | 1.71 [0.86 to 3.42] | 2.03 [0.90 to 4.58]
  M07-0241084 (Day 1, N=21,22,14,20,11,19,21,18,17) | 3.68 [2.07 to 6.54] | 4.2 [2.25 to 7.85] | 2.28 [1.16 to 4.48] | 2.36 [1.51 to 3.70] | 4.1 [1.89 to 8.90] | 7.35 [3.82 to 14] | 2.08 [1.26 to 3.42] | 2.15 [1.14 to 4.05] | 3.5 [1.57 to 7.80]
  M07-0241084 (Day 30, N=21,22,16,20,11,19,21,18,16) | 59 [36 to 98] | 4.37 [2.29 to 8.31] | 36 [20 to 64] | 2.2 [1.38 to 3.49] | 68 [33 to 142] | 66 [35 to 124] | 3.26 [1.75 to 6.06] | 2.24 [1.14 to 4.38] | 4.57 [1.48 to 14]
  M07-0241084 (Day 365,N=21,22,16,20,11,19,21,18,17) | 7.96 [4.60 to 14] | 3.28 [2.16 to 4.97] | 4.09 [2.30 to 7.25] | 2.04 [1.43 to 2.92] | 10 [4.51 to 24] | 11 [6.35 to 18] | 2.45 [1.59 to 3.79] | 1.91 [1.14 to 3.23] | 3.92 [1.90 to 8.07]
  M14459 (Day 1, N=21,22,14,20,11,20,21,18,17) | 2.69 [1.51 to 4.78] | 2.94 [1.77 to 4.89] | 1.54 [0.90 to 2.63] | 2.01 [1.40 to 2.88] | 3.11 [1.74 to 5.56] | 3.37 [1.95 to 5.81] | 1.85 [1.13 to 3.04] | 1.48 [1.03 to 2.13] | 2.55 [1.37 to 4.77]
  M14459 (Day 30, N=21,22,16,20,11,20,20,18,16) | 39 [21 to 70] | 2.31 [1.39 to 3.82] | 20 [10 to 39] | 2.03 [1.38 to 2.98] | 56 [27 to 117] | 35 [21 to 60] | 3.44 [2.05 to 5.75] | 2.71 [1.56 to 4.70] | 3.05 [1.05 to 8.83]
  M14459 (Day 365, N=21,22,16,20,11,20,21,18,17) | 7.19 [3.89 to 13] | 1.67 [1.07 to 2.60] | 2.94 [1.49 to 5.80] | 1.47 [1.07 to 2.03] | 11 [4.41 to 28] | 7.12 [3.59 to 14] | 2.09 [1.33 to 3.29] | 1.38 [0.98 to 1.93] | 2.17 [1.07 to 4.41]
  NZ98/254 (Day 1, N=21,22,14,20,11,19,21,18,17) | 1.73 [1.06 to 2.81] | 2.34 [1.33 to 4.10] | 1.34 [0.94 to 1.93] | 1.48 [1.01 to 2.17] | 1.72 [0.99 to 2.98] | 2.24 [1.20 to 4.17] | 1.18 [0.84 to 1.66] | 1.19 [0.90 to 1.58] | 1.13 [0.94 to 1.37]
  NZ98/254 (Day 30, N=21,22,16,20,11,19,21,18,16) | 32 [19 to 52] | 2.23 [1.25 to 3.99] | 15 [5.93 to 36] | 1.75 [0.98 to 3.14] | 17 [6.22 to 45] | 28 [17 to 47] | 2.48 [1.31 to 4.69] | 1.62 [0.96 to 2.74] | 1.73 [0.77 to 3.90]
  NZ98/254 (Day 365, N=21,22,16,20,11,19,21,18,17) | 3.49 [2.12 to 5.74] | 1.71 [1.14 to 2.57] | 2.67 [1.27 to 5.61] | 1.23 [0.90 to 1.69] | 3.28 [1.66 to 6.49] | 3.77 [1.98 to 7.18] | 1.65 [1.04 to 2.61] | 1.19 [0.91 to 1.54] | 1.28 [0.85 to 1.92]

22. Secondary Outcome: 22. Percentage of Subjects With HT-hSBA Titer ≥ 1:8 to N. Meningitidis Serogroups A,C,W,Y at 12 Months After Booster Vaccination.
Description: Percentage of subjects with HT-hSBA titer ≥ 1:8 to N. meningitidis serogroups A,C,W,Y at Day 1, Day 30 (one month) and Day 365 (12 months) after the administration of MenABCWY booster vaccination in this study.
Time Frame: Day 1, Day 30 and Day 365
Population: as for outcome 15
Measure: Number (95% Confidence Interval); unit: Percentages of Subjects
Arm/Group | 2OMV_OMV | 2OMV_Pbo | 2qOMV_qOMV | 2qOMV_Pbo | 2B_OMV | 2B_qOMV | 1M_OMV | 1M_qOMV | 1M_Pbo
Number analyzed (Participants) | 21 | 22 | 16 | 20 | 11 | 20 | 20 | 18 | 17
Percentages of Subjects
  Men A (Day 1, N= 21,22,15,20,10,20,20,17,17) | 38 [18.1 to 61.6] | 18 [5.2 to 40.3] | 20 [4.3 to 48.1] | 30 [11.9 to 54.3] | 30 [6.7 to 65.2] | 35 [15.4 to 59.2] | 45 [23.1 to 68.5] | 12 [1.5 to 36.4] | 41 [18.4 to 67.1]
  Men A (Day 30, N= 21,22,15,19,10,20,18,16,16) | 100 [83.9 to 100] | 32 [13.9 to 54.9] | 100 [78.2 to 100] | 26 [9.1 to 51.2] | 100 [69.2 to 100] | 95 [75.1 to 99.87] | 100 [81.5 to 100] | 94 [69.8 to 99.84] | 44 [19.8 to 70.1]
  Men A (Day 365, N= 21,22,16,20,10,20,20,18,17) | 67 [43 to 85.4] | 23 [7.8 to 45.4] | 88 [61.7 to 98.4] | 25 [8.7 to 49.1] | 90 [55.5 to 99.75] | 85 [62.1 to 96.8] | 85 [62.1 to 96.8] | 50 [26 to 74] | 35 [14.2 to 61.7]
  Men C (Day 1, N= 20,19,14,20,11,19,19,18,16) | 65 [40.8 to 84.6] | 68 [43.4 to 87.4] | 71 [41.9 to 91.6] | 65 [40.8 to 84.6] | 36 [10.9 to 69.2] | 58 [33.5 to 79.7] | 58 [33.5 to 79.7] | 50 [26 to 74] | 75 [47.6 to 92.7]
  Men C (Day 30, N= 17,20,10,20,7,14,19,17,16) | 100 [80.5 to 100] | 65 [40.8 to 84.6] | 100 [69.2 to 100] | 55 [31.5 to 76.9] | 100 [59 to 100] | 100 [76.8 to 100] | 100 [82.4 to 100] | 88 [63.6 to 98.5] | 69 [41.3 to 89]
  Men C (Day 365, N= 21,21,16,20,11,19,19,18,17) | 100 [83.9 to 100] | 62 [38.4 to 81.9] | 100 [79.4 to 100] | 50 [27.2 to 72.8] | 82 [48.2 to 97.7] | 95 [74 to 99.87] | 100 [82.4 to 100] | 89 [65.3 to 98.6] | 65 [38.3 to 85.8]
  Men W (Day 1, 20,22,12,20,11,20,17,18,16) | 95 [75.1 to 99.87] | 95 [77.2 to 99.88] | 75 [42.8 to 94.5] | 70 [45.7 to 88.1] | 82 [48.2 to 97.7] | 75 [50.9 to 91.3] | 82 [56.6 to 96.2] | 61 [35.7 to 82.7] | 56 [29.9 to 80.2]
  Men W (Day 30, N= 18,22,15,19,11,18,17,16,14) | 100 [81.5 to 100] | 86 [65.1 to 97.1] | 100 [78.2 to 100] | 74 [48.8 to 90.9] | 100 [71.5 to 100] | 100 [81.5 to 100] | 100 [80.5 to 100] | 100 [79.4 to 100] | 57 [28.9 to 82.3]
  Men W (Day 365, N= 21,22,16,20,11,20,19,18,17) | 100 [83.9 to 100] | 82 [59.7 to 94.8] | 100 [79.4 to 100] | 65 [40.8 to 84.6] | 91 [58.7 to 99.77] | 100 [83.2 to 100] | 100 [82.4 to 100] | 100 [81.5 to 100] | 65 [38.3 to 85.8]
  Men Y (Day 1, N= 21,21,14,20,11,18,20,18,17) | 62 [38.4 to 81.9] | 62 [38.4 to 81.9] | 71 [41.9 to 91.6] | 40 [19.1 to 63.9] | 36 [10.9 to 69.2] | 11 [1.4 to 34.7] | 55 [31.5 to 76.9] | 44 [21.5 to 69.2] | 41 [18.4 to 67.1]
  Men Y (Day 30, N= 21,21,15,20,11,18,20,17,16) | 100 [83.9 to 100] | 57 [34 to 78.2] | 100 [78.2 to 100] | 40 [19.1 to 63.9] | 82 [48.2 to 97.7] | 83 [58.6 to 96.4] | 100 [83.2 to 100] | 100 [80.5 to 100] | 38 [15.2 to 64.6]
  Men Y (Day 365, N= 21,21,16,20,11,18,20,18,17) | 95 [76.2 to 99.88] | 52 [29.8 to 74.3] | 100 [79.4 to 100] | 40 [19.1 to 63.9] | 45 [16.7 to 76.6] | 72 [46.5 to 90.3] | 100 [83.2 to 100] | 89 [65.3 to 98.6] | 47 [23 to 72.2]

23. Secondary Outcome: 23. Number of Subjects With Solicited Local and Systemic Adverse Events Following Booster Vaccination in This Study.
Description: Number of subjects reporting solicited local and systemic adverse events after receiving a booster dose of MenABCWY vaccine or placebo. the below reported events are Erythema- Injection site erythema, Induration- Injection site induration, Pain-injection site pain, Arthralgia, Chills, Fatigue, Headache, Loss of Appetite, Myalgia, Nausea, Rash, Fever, Prevention- Prevention of Pain and/or Fever, Treatment- Treatment of Pain and/or Fever and Analgesic/Antipyr.: use of Analgesic/Antipyretics in pain and fever.
Time Frame: From day 1 (6 hours) through day 7 after any vaccination
Population: Analysis was done on the Solicited Safety Set, i.e. all exposed subjects who provide post vaccination solicited adverse event data.
Measure: Number; unit: Participants
Arm/Group | 2OMV_OMV | 2OMV_Pbo | 2qOMV_qOMV | 2qOMV_Pbo | 2B_OMV | 2B_qOMV | 2B_Pbo | 1M_OMV | 1M_qOMV | 1M_Pbo | Total
Number analyzed (Participants) | 26 | 24 | 17 | 23 | 11 | 21 | 6 | 21 | 19 | 19 | 187
Participants
  Any AEs (N=26,24,17,23,11,21,6,21,19,19,187) | 23 | 10 | 15 | 13 | 11 | 18 | 2 | 20 | 17 | 8 | 137
  Any Local (N=26,24,17,23,11,21,6,21,19,19,187) | 23 | 7 | 15 | 8 | 11 | 18 | 1 | 19 | 17 | 5 | 124
  Erythema (N=26,23,17,23,11,21,6,21,19,19,186) | 11 | 2 | 7 | 3 | 6 | 7 | 0 | 6 | 9 | 2 | 53
  Induration (N=26,23,17,23,11,21,6,21,19,18,185) | 7 | 2 | 5 | 2 | 9 | 6 | 0 | 11 | 9 | 1 | 52
  Pain (N=26,24,17,23,11,21,6,21,19,19,187) | 20 | 6 | 14 | 7 | 11 | 17 | 1 | 19 | 17 | 4 | 116
  Any Systemic (N=26,24,17,23,11,21,6,21,19,19,187) | 12 | 9 | 12 | 6 | 6 | 10 | 1 | 15 | 10 | 5 | 86
  Arthralgia(N=25,23,17,23,10,21,6,21,19,19,184) | 3 | 2 | 3 | 1 | 0 | 2 | 0 | 4 | 2 | 3 | 20
  Chills(N=26,23,17,23,11,21,6,21,19,19,186) | 3 | 1 | 0 | 0 | 1 | 2 | 0 | 5 | 1 | 1 | 14
  Fatigue(N=26,23,17,23,11,21,6,21,19,19,186) | 9 | 6 | 8 | 2 | 5 | 8 | 0 | 11 | 6 | 5 | 60
  Headache(N=26,23,17,23,11,21,6,21,19,19,186) | 7 | 6 | 8 | 3 | 5 | 4 | 1 | 12 | 5 | 2 | 53
  Loss ofAppetite(N=26,23,17,23,11,21,6,21,19,19,186 | 2 | 1 | 4 | 2 | 1 | 3 | 0 | 8 | 3 | 2 | 26
  Myalgia(N=26,23,17,23,10,21,6,21,19,19,185) | 6 | 2 | 5 | 0 | 1 | 4 | 0 | 8 | 4 | 1 | 31
  Nausea(N=26,23,17,23,11,21,6,21,19,19,186) | 0 | 2 | 3 | 1 | 3 | 5 | 0 | 4 | 5 | 1 | 24
  Rash (N=26,23,17,23,11,21,6,21,18,19,185) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 2 | 0 | 5
  Fever >38 °C (N=25,24,17,23,11,21,6,21,19,18,185) | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 3
  Prevention (N=25,23,17,23,11,21,6,21,19,19,185) | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
  Treatment (N=25,23,17,23,11,21,6,21,19,19,185) | 2 | 1 | 3 | 2 | 1 | 5 | 0 | 6 | 2 | 0 | 22
  Analgesic/Antipyr. Pain (N=0,0,1,0,0,0,0,0,0,0,1) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Analgesic/Antipyr. Fever (N=0,0,1,0,0,0,0,0,0,0,1) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

24. Secondary Outcome: 24. Number of Subjects With Unsolicited (Any AEs and Possibly Related AEs) Following Booster Vaccination in This Study.
Description: Number of subjects reporting unsolicited AEs (any AEs and at least possibly related AEs) after receiving a booster dose of MenABCWY vaccine or placebo from Day 1 to Day 30.
  Analysis was done on the Unsolicited Safety Set. All subjects in the exposed population who provided information about post-vaccination AEs or safety records at Day 30.
Time Frame: Day 1 through Day 30
Population: Analysis was done on the Unsolicited Safety Set. All subjects in the exposed population who provided information about post-vaccination AEs or safety records at Day 30.
Measure: Number; unit: Participants
Arm/Group | 2OMV_OMV | 2OMV_Pbo | 2qOMV_qOMV | 2qOMV_Pbo | 2B_OMV | 2B_qOMV | 2B_Pbo | 1M_OMV | 1M_qOMV | 1M_Pbo
Number analyzed (Participants) | 26 | 24 | 17 | 23 | 11 | 21 | 6 | 21 | 19 | 19
Participants
  Any AEs | 6 | 4 | 5 | 2 | 3 | 7 | 1 | 6 | 5 | 4
  At least possibly related | 3 | 1 | 3 | 0 | 2 | 3 | 0 | 2 | 3 | 0

25. Secondary Outcome: 25. Number of Subjects With Unsolicited Adverse Events Following Booster Vaccination in This Study.
Description: Number of subjects reporting any serious unsolicited AEs (SAEs), possibly related SAEs, medically attended AEs, unsolicited AEs leading to withdrawal and deaths after receiving a booster dose of MenABCWY vaccine or placebo, are reported for the entire study period.
Time Frame: Day 1 to Day 365
Population: as for outcome 24
Measure: Number; unit: Participants
Arm/Group | 2OMV_OMV | 2OMV_Pbo | 2qOMV_qOMV | 2qOMV_Pbo | 2B_OMV | 2B_qOMV | 2B_Pbo | 1M_OMV | 1M_qOMV | 1M_Pbo
Number analyzed (Participants) | 26 | 24 | 17 | 23 | 11 | 21 | 6 | 21 | 19 | 19
Participants
  Any SAEs | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 1 | 1
  At Least Possibly related SAEs | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  NOCD | 0 | 3 | 2 | 0 | 0 | 1 | 0 | 1 | 1 | 1
  Medically attended AEs | 12 | 10 | 12 | 9 | 6 | 9 | 1 | 13 | 11 | 11
  AEs leading to withdrawal | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Deaths | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

26. Secondary Outcome: 26. Number of Subjects With Unsolicited Adverse Leading to New Onset Chronic Disease (NOCD) Before Study Vaccination.
Description: Number of subjects reporting New Onset Chronic Disease (NOCD),from the end of the primary parental study V102_03 (NCT01272180) up to Day 1 visit in V102_03E1 study, is reported. (Any NOCD AEs: NOCD V102_03 (NCT01272180) vs. NOCD- Day 1, V102_03E1)
Time Frame: From primary parent study completion up to Day 1 in this study.
Population: Analysis was done on the all enrolled set population. All screened subjects who have been enrolled (ie, attended the first clinic visit and received a subject ID).
Measure: Number; unit: Participants
Arm/Group | 2OMV_OMV | 2OMV_Pbo | 2qOMV_qOMV | 2qOMV_Pbo | 2B_OMV | 2B_qOMV | 2B_Pbo | 1M_OMV | 1M_qOMV | 1M_Pbo
Number analyzed (Participants) | 26 | 25 | 17 | 24 | 11 | 21 | 7 | 21 | 19 | 19
Participants | 2 | 4 | 0 | 1 | 0 | 2 | 1 | 2 | 2 | 1

ADVERSE EVENTS:
Time Frame: Solicited adverse events (AEs) between Day 1 (from 30 minutes) to Day 7; any unsolicited AE from Day 1 (from 30 minutes) to Day 30 and serious AE, medically attended AE, AE leading to withdrawal, death and NOCD from Day 1 to Day 365.
Description: Safety analysis was conducted on the solicited and unsolicited safety set cohorts that included only the exposed subjects who provided solicited adverse event data and post-vaccination AE data, respectively.
Groups:
- Total: Total
Arm/Group | 2OMV_OMV | 2OMV_Pbo | 2qOMV_qOMV | 2qOMV_Pbo | 2B_OMV | 2B_qOMV | 2B_Pbo | 1M_OMV | 1M_qOMV | 1M_Pbo | Total
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/24 | 1/17 | 1/23 | 0/11 | 1/21 | 0/6 | 0/21 | 1/19 | 1/19 | 5/188
Other Adverse Events (participants affected / at risk) | 25/26 | 16/24 | 16/17 | 15/23 | 11/11 | 19/21 | 4/6 | 20/21 | 17/19 | 15/19 | 158/188
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 2OMV_OMV (N=26) | 2OMV_Pbo (N=24) | 2qOMV_qOMV (N=17) | 2qOMV_Pbo (N=23) | 2B_OMV (N=11) | 2B_qOMV (N=21) | 2B_Pbo (N=6) | 1M_OMV (N=21) | 1M_qOMV (N=19) | 1M_Pbo (N=19) | Total (N=188)
Appendicitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Facial bones fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Limb injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Syncope (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 2OMV_OMV (N=26) | 2OMV_Pbo (N=24) | 2qOMV_qOMV (N=17) | 2qOMV_Pbo (N=23) | 2B_OMV (N=11) | 2B_qOMV (N=21) | 2B_Pbo (N=6) | 1M_OMV (N=21) | 1M_qOMV (N=19) | 1M_Pbo (N=19) | Total (N=188)
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Myopia (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2
Photophobia (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Nausea (Gastrointestinal disorders) | 1 | 2 | 3 | 1 | 3 | 5 | 0 | 4 | 5 | 1 | 25
Tooth impacted (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Chills (General disorders) | 3 | 1 | 0 | 0 | 1 | 2 | 0 | 6 | 1 | 1 | 15
Fatigue (General disorders) | 9 | 8 | 8 | 2 | 5 | 8 | 0 | 11 | 6 | 5 | 62
Induration (General disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2
Injection site erythema (General disorders) | 11 | 2 | 7 | 3 | 7 | 7 | 0 | 7 | 9 | 2 | 55
Injection site induration (General disorders) | 7 | 2 | 6 | 3 | 10 | 7 | 0 | 11 | 9 | 1 | 56
Injection site pain (General disorders) | 21 | 7 | 14 | 7 | 11 | 18 | 1 | 19 | 17 | 6 | 121
Injection site pruritus (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2
Pyrexia (General disorders) | 2 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 4
Vaccination site erythema (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vaccination site pain (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Acute sinusitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Bronchitis (Infections and infestations) | 0 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 5
Conjunctivitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 3
Croup infectious (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Herpes virus infection (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 2
Influenza (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 3
Laryngitis (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Lice infestation (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Nasopharyngitis (Infections and infestations) | 0 | 2 | 0 | 1 | 1 | 2 | 0 | 1 | 0 | 1 | 8
Onychomycosis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Otitis media (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Pharyngitis (Infections and infestations) | 1 | 2 | 2 | 0 | 1 | 1 | 0 | 2 | 0 | 1 | 10
Pharyngitis streptococcal (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 4
Pneumonia (Infections and infestations) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 3
Pneumonia mycoplasmal (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Sinusitis (Infections and infestations) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 3
Tonsillitis (Infections and infestations) | 2 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 4
Tooth abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 2 | 1 | 1 | 1 | 0 | 2 | 2 | 1 | 10
Viral infection (Infections and infestations) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Viral pharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 3
Concussion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 2
Head injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Limb injury (Injury, poisoning and procedural complications) | 2 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 6
Post vaccination syndrome (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Blood iron decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Body temperature increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Abnormal weight gain (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 2 | 1 | 4 | 2 | 1 | 3 | 1 | 8 | 4 | 2 | 28
Obesity (Metabolism and nutrition disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 2 | 3 | 1 | 0 | 2 | 0 | 4 | 2 | 3 | 21
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 6 | 2 | 5 | 0 | 1 | 4 | 0 | 8 | 4 | 1 | 31
Myositis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Scoliosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Temporomandibular joint syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Dizziness postural (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 8 | 6 | 8 | 3 | 5 | 4 | 1 | 14 | 5 | 2 | 56
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Proteinuria (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Breast mass (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 3
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 5
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 2
Acne (Skin and subcutaneous tissue disorders) | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 5
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 2
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 3 | 2 | 0 | 7
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 2
Essential hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No